CLINICAL TRIAL: NCT01587898
Title: A Four-week Phase IIa, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multi-center Study to Evaluate the Safety, Efficacy and Pharmacokinetics of GSK1278863 in Subjects With Anemia Associated With Chronic Kidney Disease Who Are Not Taking Recombinant Human Erythropoietin and Are Not Undergoing Dialysis
Brief Title: 4 Week Correction Study in Subjects With Anemia Associated With Chronic Kidney Disease Who Are Not Undergoing Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116581
Record Dates: First submitted 2012-04-19; First posted 2012-04-30 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-08

CONDITIONS: Anaemia
Keywords: Anemia; Prolyl hydroxylase inhibitor; Hemoglobin; Chronic kidney disease; pharmacokinetics; recombinant human erythropoietin; GSK1278863
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — GSK1278863

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.5mg GSK1278863 (Experimental): Once daily
  Interventions: Drug: GSK1278863
- 2mg GSK1278863 (Experimental): Once daily
  Interventions: Drug: GSK1278863
- 5mg GSK1278863 (Experimental): Once daily
  Interventions: Drug: GSK1278863
- Placebo (Experimental): Once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GSK1278863 — Tablet
  Arms: 0.5mg GSK1278863; 2mg GSK1278863; 5mg GSK1278863
Other: Placebo — Tablet
  Arms: Placebo

SUMMARY:
This is a four-week Phase IIa, randomized, double-blind, placebo-controlled, parallel-group, multi-center study to evaluate the safety, efficacy and pharmacokinetics of GSK1278863 in approximately 68 subjects with anemia associated with chronic kidney disease who are not taking rhEPO and are not undergoing dialysis. The range of Hgb values for study eligibility is 8.5-11.0 g/dL. Eligible subjects will be randomized in equal proportions to receive once daily (QD) placebo or GSK1278863 0.5 mg, 2 mg or 5 mg in a double-blind fashion.

DETAILED DESCRIPTION:
This is a four-week Phase IIa, randomized, double-blind, placebo-controlled, parallel-group, multi-center study to evaluate the safety, efficacy and pharmacokinetics of GSK1278863 in approximately 68 subjects with anemia associated with chronic kidney disease who are not taking rhEPO and are not undergoing dialysis. The study consists of a screening phase of up to 2 weeks, a 4-week treatment phase and a 2-week follow-up phase. The range of Hgb values for study eligibility is 8.5-11.0 g/dL. Eligible subjects will be randomized in equal proportions to receive once daily (QD) placebo or GSK1278863 0.5 mg, 2 mg or 5 mg in a double-blind fashion. Study treatment will be stopped if Hgb values fall outside of the range pre-specified in the protocol.

This study aims to estimate the relationship between dose of GSK1278863 and Hgb response for correcting anemia in non-dialysis subjects with CKD who are not taking rhEPO (NDD). In addition, the study will characterize the effect of GSK1278863 on various pharmacokinetic/pharmacodynamic (PK/PD) markers, and will investigate the safety and tolerability of GSK1278863.

An early interim analysis of the Hgb data is planned after approximately 20 subjects from cohort 1 have completed 3 weeks of treatment. Depending upon the interim findings, a second cohort of subjects may be added to investigate an additional GSK1278863 dose arm. Recruitment to the first cohort will continue during the interim analysis.

A second interim analysis is planned after approximately 48 subjects from cohort 1 have completed 4 weeks treatment. The purpose of this interim is three-fold, to investigate whether a second cohort of subjects may be added, to facilitate early development of dose-response and PK/PD statistical models, and to generate interim results to facilitate design and dosing decisions for the next trial.

Subject completion is defined as completion of all study phases including the follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

1. Age and weight: >/= 18 years of age and >/= 45 kg.
2. Not routinely undergoing dialysis, regardless of the modality (either hemodialysis or peritoneal dialysis) or dialysis planned during the time the subject would be enrolled in the study.
3. No current or prior rhEPO use within the past 7 weeks; e.g., epoetins (or their biosimilars), darbepoetin, Mircera (methoxy polyethylene glycol epoetin beta), peginesatide or their biosimilars..
4. KDOQI CKD stages 3/4/5 defined by eGFR using the Modification of Diet for Renal Disease (MDRD).
5. Hgb: Hgb concentrations 8.5-11.0 g/dL (inclusive) as outlined in Section 4.2.
6. Vitamin B12: Above the lower limit of the reference range (may rescreen in 2 months).
7. Folate: >/=2.0 ng/mL at Screening. May rescreen in a month.
8. Ferritin: >/=40 ng/mL with the absence of microcytic or hypochromic RBCs.
9. TSAT within the reference range.
10. Iron replacement therapy: Stable maintenance dose of oral iron replacement therapy, if required, that will be maintained throughout the study. NOTE: IV iron replacement therapy is not allowed the two weeks prior to Screening through the end of the study (Week 6).
11. QTc: QTcB <470 msec or QTcB <480 msec in subjects with bundle branch block obtained at Screening Visit, based on Central Reader's interpretation.
12. Females: Eligible to participate if she is of childbearing potential, and must agree to use approved contraception methods from Screening until completion of the Follow-up Visit OR of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation of hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH)>40 MIU/ml and estradiol <40 pg/ml is confirmatory]. Females on hormone replacement therapy (HRT) whose menopausal status is in doubt will be required to use one of the approved contraception methods if they wish to continue their HRT during the study. Otherwise they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most types of HRT, at least 2 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
13. Males: Must agree to use approved contraceptive methods from the time of Screening until completion of the Follow-up Visit.

Exclusion Criteria:

1. Dialysis: Planning to initiate dialysis during the study or who have a high potential for initiating dialysis during study participation.
2. Renal transplant: Renal transplant anticipated or scheduled within the study time period or subjects with a functioning renal transplant.
3. Total CPK: >5x the upper limit of the reference range.
4. HIV: Positive HIV antibody.
5. History of myocardial infarction or acute coronary syndrome within the prior 6 months.
6. History of stroke or TIAs.
7. Heart failure: Class III/IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
8. Hypertension: Poorly controlled hypertension, whether due to inadequate treatment, or lack of treatment, defined as DBP >100 mmHg or SBP>160 mmHg.
9. Thrombotic disease: History of thrombotic disease (e.g., venous thrombosis such as deep vein thrombosis or pulmonary embolism, or arterial thrombosis such as new onset or worsening limb ischemia requiring intervention), or other thrombosis related condition) within the prior 6 months.
10. Pulmonary hypertension: Known pulmonary hypertension and those at higher risk (than normally associated with CKD) for pre-existing elevation in pulmonary pressure (e.g., significant heart failure or lung disease requiring supplemental oxygen, or those with connective tissue diseases).
11. Inflammatory disease: Chronic inflammatory disease that could impact erythropoiesis (e.g., scleroderma, systemic lupus erythematosis, rheumatoid arthritis, celiac disease).
12. Hematological disease: Any hematological disease including those affecting platelets, the coagulation disorders (e.g., Protein C or S deficiency) or red blood cells (e.g. sickle cell anemia, myelodysplastic syndromes, hematological malignancy, myeloma, hemolytic anemia) or any other cause of anemia other than renal disease.
13. Liver disease: Current liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) or evidence at Screening of abnormal liver function tests [alkaline phosphatase, ALT or AST > 2.0 x upper limit of normal (ULN) or total bilirubin > 1.5 x ULN]; or other hepatic abnormalities that in the opinion of the investigator would preclude the subject from participation in the study.
14. Major surgery: Within the prior 12 weeks or planned during the study.
15. Transfusion: Blood transfusion within the prior 12 weeks or an anticipated need for blood transfusion during the study.
16. Ulcer and Active GI Bleeding: Evidence of active peptic, duodenal, or esophageal ulcer disease or active GI bleeding within the prior 12 weeks.
17. Acute infection: Clinical evidence of acute infection or history of infection requiring intravenous (IV) antibiotic therapy the eight weeks prior to Screening through Day 1 (randomization).
18. Malignancy: History of malignancy within 5 years of Screening or are receiving treatment for cancer or those with a strong family history of cancer (e.g., familial cancer disorders), with the exception of squamous cell or basal cell carcinoma of the skin that has been definitively treated.
19. Hyperparathyroidism: Clinically significant hyperparathyroidism in the opinion of the Investigator, including subjects with parathyroid hormone (PTH) values ≥600 pg/mL.
20. Eyes: History of proliferative retinopathy requiring treatment within the prior 12 months, or macular edema requiring treatment.
21. Severe reactions: History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product.
22. Drugs and supplements: Use of any prescription or non-prescription drugs or dietary supplements that are prohibited from Screening until the Follow-up Visit.
23. Androgens: New androgen therapy or changes to pre-existing androgen regimen within prior 12 weeks.
24. Prior investigational product exposure: The subject has participated in a clinical trial and has received an experimental investigational product within prior 30 days.
25. Protocol compliance: Unwillingness or inability to follow the procedures, or lifestyle and/or dietary restrictions outlined in the protocol.
26. Other conditions: Any condition which in the investigators opinion should exclude the subject from participating in the study.
27. Pregnancy and lactation: Pregnant females as determined by positive urine hCG test, OR women who are lactating at Screening or during the trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-05-17 (Actual); Primary Completion 2013-05-07 (Actual); Study Completion 2013-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (50):
- United States (41):
  - GSK Investigational Site, Azusa, California
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Chino, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, North Hollywood, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Dimas, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Yuba City, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Edgewater, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Port Charlotte, Florida
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Evanston, Illinois
  - GSK Investigational Site, Gurnee, Illinois
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Greenville, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Silverdale, Washington
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, London, Ontario
- Germany (5):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Lehrte, Lower Saxony
  - GSK Investigational Site, Demmin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Holdstock L, Meadowcroft AM, Maier R, Johnson BM, Jones D, Rastogi A, Zeig S, Lepore JJ, Cobitz AR. Four-Week Studies of Oral Hypoxia-Inducible Factor-Prolyl Hydroxylase Inhibitor GSK1278863 for Treatment of Anemia. J Am Soc Nephrol. 2016 Apr;27(4):1234-44. doi: 10.1681/ASN.2014111139. Epub 2015 Oct 22. PMID 26494831
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 116581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at Canada, Germany, and United States between 29 May 2012 and 30 May 2013. A total of 282 participants were screened, 209 were screen failures and 73 eligible participants were randomized. Entry into the study requires a target stable hemoglobin (Hgb) of 8.5-11.0 gram per deciliter (g/dL).
Pre-assignment Details: Out of the 73 randomized participants, one participant did not receive any study medication. the remaining 72 participants were included in safety population. Another one participant had no post-randomization data and was excluded from Intent-to-treat (ITT) population (71 participants).
Groups:
- Placebo: Eligible participants received two matching placebo tablets, one each from bottle A and B once daily, orally, in the morning of each dosing day with a glass of water for 4 weeks except when the participants were dosed on-site by study personnel on Day 1 and at Week 4 clinic visit.
- GSK1278863, 0.5 mg: Eligible participants received one GSK1278863 0.5 milligram (mg) tablet from bottle A and one matching placebo tablets from bottle B once daily, orally, in the morning of each dosing day with a glass of water for 4 weeks except when the participants were dosed on-site by study personnel on Day 1 and at Week 4 clinic visit.
- GSK1278863, 2 mg: Eligible participants received one GSK1278863 2 mg tablet from bottle A and one matching placebo tablets from bottle B once daily, orally, in the morning of each dosing day with a glass of water for 4 weeks except when the participants were dosed on-site by study personnel on Day 1 and at Week 4 clinic visit.
- GSK1278863, 5 mg: Eligible participants received one GSK1278863 5 mg tablet from bottle B and one matching placebo tablets from bottle A once daily, orally, in the morning of each dosing day with a glass of water for 4 weeks except when the participants were dosed on-site by study personnel on Day 1 and at Week 4 clinic visit.
Period: Overall Study
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Started | 18 | 17 | 18 | 19
Completed | 14 | 12 | 16 | 17
Not Completed | 4 | 5 | 2 | 2
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Not completed — Met haemoglobin stopping criteria | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK1278863, 0.5 mg: Eligible participants received one GSK1278863 0.5 mg tablet from bottle A and one matching placebo tablets from bottle B once daily, orally, in the morning of each dosing day with a glass of water for 4 weeks except when the participants were dosed on-site by study personnel on Day 1 and at Week 4 clinic visit.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg | Total
Number analyzed (Participants) | 18 | 17 | 18 | 19 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.2 (11.00) | 66.6 (11.73) | 66.9 (11.45) | 71.3 (11.26) | 68.6 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 10 | 16 | 52
  Male | 4 | 5 | 8 | 3 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 4 | 5 | 20
  Not Hispanic or Latino | 12 | 12 | 14 | 14 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Modeled Hgb Change From Baseline Over 4 Weeks of Treatment
Description: Modeled Hgb change from baseline over 4 weeks was derived using a random coefficient mixed effects linear regression model. The model included fixed effects for baseline Hgb, treatment and a treatment by day interaction. Random effects was fitted in the intercept and the slope over time. All data up until investigational product discontinuation was included for Hgb efficacy evaluable participants; where efficacy evaluable was defined as having a baseline and at least 2 on-treatment Hgb assessments. Baseline was the average of Week -2 , Week -1 and Day 1 visits. The change from Baseline was calculated by subtracting the Baseline value from the individual post-dose visit values.
Time Frame: Baseline (average of Week -2, -1 and Day 1) and Week 4
Population: The ITT population comprised of all randomized participants who received at least one dose of study medication, and had a baseline and at least one corresponding on treatment laboratory assessment. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: gram per decilitre (g/dL)
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 13 | 17 | 18
gram per decilitre (g/dL) | -0.148 (0.1925) | 0.132 (0.2200) | 0.463 (0.2173) | 1.010 (0.2614)
Statistical Analysis 1: Comparison: Placebo vs GSK1278863, 0.5 mg vs GSK1278863, 2 mg vs GSK1278863, 5 mg; Subgroup: Baseline Hgb; Test type: Superiority or Other; p = 0.5888, Mixed effects linear regression model; The modeled Hgb change from baseline over 4 weeks was derived using a random coefficient mixed effects linear regression model
Statistical Analysis 2: Comparison: Placebo vs GSK1278863, 0.5 mg vs GSK1278863, 2 mg vs GSK1278863, 5 mg; Subgroup: Baseline Weight; Test type: Superiority or Other; p = 0.6600, Mixed effects linear regression model; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs GSK1278863, 0.5 mg vs GSK1278863, 2 mg vs GSK1278863, 5 mg; Subgroup: Baseline estimated glomerular filtration rate (eGFR); Test type: Superiority or Other; p = 0.7999, Mixed effects linear regression model; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs GSK1278863, 0.5 mg vs GSK1278863, 2 mg vs GSK1278863, 5 mg; Covariate: Ethnicity; Test type: Superiority or Other; p = 0.2092, Mixed effects linear regression model; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs GSK1278863, 0.5 mg vs GSK1278863, 2 mg vs GSK1278863, 5 mg; Covariate: Geographic Ancestry; Test type: Superiority or Other; p = 0.9996, Mixed effects linear regression model; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs GSK1278863, 0.5 mg vs GSK1278863, 2 mg vs GSK1278863, 5 mg; Covariate: Sex; Test type: Superiority or Other; p = 0.7002, Mixed effects linear regression model; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs GSK1278863, 0.5 mg vs GSK1278863, 2 mg vs GSK1278863, 5 mg; Covariate: Age; Test type: Superiority or Other; p = 0.5536, Mixed effects linear regression model; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs GSK1278863, 0.5 mg vs GSK1278863, 2 mg vs GSK1278863, 5 mg; Co-administration with food; Test type: Superiority or Other; p = 0.0085, Mixed effects linear regression model; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs GSK1278863, 0.5 mg vs GSK1278863, 2 mg vs GSK1278863, 5 mg; Covariate: Diabetic; Test type: Superiority or Other; p = 0.0021, Mixed effects linear regression model; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs GSK1278863, 0.5 mg vs GSK1278863, 2 mg vs GSK1278863, 5 mg; Covariate: Region; Test type: Superiority or Other; p = 0.2194, Mixed effects linear regression model; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Model-Adjusted Maximum Hgb Changes Over 4 Weeks
Description: Maximum Hgb change over 4 weeks was analyzed using an ANCOVA model with terms included for treatment and baseline Hgb value. Least square mean estimates and 95% CI for each treatment group were reported. Baseline was the average of Week -2 , Week -1 and Day 1 visits. The change from Baseline was calculated by subtracting the baseline value from the individual post-dose visit values.
Time Frame: Baseline (average of Week -2 , -1 and Day 1 visits) and 4 weeks
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
g/dL | 0.153 (0.1476) | 0.137 (0.1609) | 0.474 (0.1532) | 1.069 (0.1527)

3. Secondary Outcome: Number of Participants Achieving an Increase of 0.5, 1.0, 1.5 and 2.0 g/dL in Hgb
Description: Number of participants achieving an increase of 0.5, 1.0, 1.5 and 2.0 g/dL in Hgb from baseline were reported. Entry into the study required a target stable Hgb of 8.5-11.0 g/dL. A stable Hgb value was confirmed from three Hgb values taken during the screening period at Week -2, Week -1 and Day 1 (randomization). The average of these three values was used for Baseline Hgb.
Time Frame: Up to 4 weeks
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
Participants
  Decrease/increase of < 0.5 g/dL | 16 | 12 | 12 | 4
  Increase of >=0.5 g/dL | 3 | 4 | 6 | 14
  Increase of >=1 g/dL | 1 | 1 | 2 | 9
  Increase of >=1.5 g/dL | 0 | 0 | 0 | 5
  Increase of >=2 g/dL | 0 | 0 | 0 | 1

4. Secondary Outcome: Percentage of Participants Achieving an Increase of 0.5, 1.0, 1.5 and 2.0 g/dL in Hgb
Description: Percentage of participants achieving an increase of 0.5, 1.0, 1.5 and 2.0 g/dL in Hgb from baseline were reported. Entry into the study requires a target stable Hgb of 8.5-11.0 g/dL. A stable Hgb value was confirmed from three Hgb values taken during the screening period at Week -2, Week -1 and Day 1 (randomization). The average of these three values was used for Baseline Hgb.
Time Frame: Up to 4 weeks
Population: ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
Percentage of participants
  Decrease/increase of < 0.5 g/dL | 84 | 75 | 67 | 22
  Increase of >=0.5 g/dL | 16 | 25 | 33 | 78
  Increase of >=1 g/dL | 5 | 6 | 11 | 50
  Increase of >=1.5 g/dL | 0 | 0 | 0 | 28
  Increase of >=2 g/dL | 0 | 0 | 0 | 6

5. Secondary Outcome: Number of Participants Who Reached Hgb Stopping Criteria
Description: The Hgb stopping criteria was defined as reaching to value <8.0 g/dL, >=8.0 - <13.0 (>= 2g/dL absolute Hgb change over 1 week ) or >=13.0 g/dL. The number of participants who reached the Hgb stopping criteria of Hgb concentration were presented.
Time Frame: Up to Week 4
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
Participants
  <8.0 | 0 | 0 | 1 | 0
  >=8.0-<13.0 and >=2.0 decrease | 1 | 0 | 0 | 0
  >=8.0-<13.0 and >=2.0 increase | 0 | 1 | 1 | 0

6. Secondary Outcome: Change From Baseline in Hepcidin at Week 2 and Week 4
Description: Blood samples for hepcidin were collected at Day 1 (pre-dose), Week 2 (approximately between 4 to 8 h) and Week 4 (pre-dose). Hepcidin is a regulator of iron metabolism. Baseline was the last pre-dose value on Day 1. The change from Baseline was calculated by subtracting the Baseline value from the individual post-dose visit values. Where hepcidin values were missing because the value was below the quantification limit (BQL), the BQL value was imputed.
Time Frame: Baseline (Pre-dose on Day 1), Week 2 and 4
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per Litre (mcg/L)
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
Microgram per Litre (mcg/L)
  Week 2: number analyzed (Participants) | 17 | 13 | 16 | 18
  Week 2 | 10.19 (88.535) | -23.46 (58.809) | -75.24 (88.862) | -120.31 (113.653)
  Week 4: number analyzed (Participants) | 15 | 10 | 15 | 16
  Week 4 | -2.62 (96.176) | -22.16 (120.138) | -77.34 (96.843) | -143.09 (119.617)

7. Secondary Outcome: Change From Baseline in Ferritin at Week 2 and Week 4
Description: Baseline was the Day 1 pre-dose value. The change from Baseline was calculated by subtracting the Baseline value from the individual post-dose visit values.
Time Frame: Baseline (Day 1 Pre-dose), Week 2 and 4
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
mcg/L
  Week 2: number analyzed (Participants) | 18 | 14 | 18 | 18
  Week 2 | 2.6 (50.49) | -20.0 (40.02) | -38.6 (70.20) | -58.8 (58.20)
  Week 4: number analyzed (Participants) | 15 | 12 | 17 | 17
  Week 4 | -24.3 (38.61) | -35.8 (54.68) | -8.2 (268.77) | -101.8 (91.07)

8. Secondary Outcome: Change From Baseline in Transferrin at Week 2 and Week 4
Description: as for outcome 7
Time Frame: Baseline (Day 1 Pre-dose), Week 2 and 4
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per litre (G/L)
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
Grams per litre (G/L)
  Week 2: number analyzed (Participants) | 17 | 14 | 18 | 18
  Week 2 | -0.017 (0.2551) | -0.100 (0.2194) | 0.153 (0.4556) | 0.141 (0.7335)
  Week 4: number analyzed (Participants) | 15 | 12 | 17 | 17
  Week 4 | 0.011 (0.2646) | 0.028 (0.2743) | 0.294 (0.3442) | 0.388 (0.3550)

9. Secondary Outcome: Change From Baseline in Transferrin Saturation at Week 2 and Week 4
Description: Transferrin saturation was measured as a percentage, and is the ratio of serum iron and total iron-binding capacity, multiplied by 100. Baseline value for transferrin saturation was the pre-dose value on Day 1. The change from Baseline was calculated by subtracting the Baseline value from the individual post-dose visit values.
Time Frame: Baseline (Day 1 Pre-dose), Week 2 and 4
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of transferrin saturation
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
Percentage of transferrin saturation
  Week 2: number analyzed (Participants) | 18 | 14 | 17 | 17
  Week 2 | 0.7 (7.18) | -1.5 (4.16) | -3.7 (4.59) | -2.1 (6.51)
  Week 4: number analyzed (Participants) | 15 | 12 | 17 | 17
  Week 4 | 1.5 (6.08) | -3.1 (4.85) | -2.6 (6.18) | -3.4 (11.27)

10. Secondary Outcome: Change From Baseline in Total Iron Binding Capacity at Week 2 and Week 4
Description: Total iron-binding capacity is a medical laboratory test that measures the blood's capacity to bind iron with transferrin. Baseline was the Day 1 pre-dose value. The change from Baseline was calculated by subtracting the Baseline value from the individual post-dose visit values.
Time Frame: Baseline (Day 1 Pre-dose), Week 2 and 4
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromol per litre (micromol/L)
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
Micromol per litre (micromol/L)
  Week 2: number analyzed (Participants) | 18 | 14 | 17 | 17
  Week 2 | 0.6 (5.63) | -1.6 (5.08) | 2.9 (3.30) | 5.9 (6.85)
  Week 4: number analyzed (Participants) | 15 | 12 | 17 | 17
  Week 4 | -0.5 (3.72) | 0.3 (6.34) | 5.1 (4.12) | 8.3 (5.54)

11. Secondary Outcome: Change From Baseline in Total Iron at Week 2 and Week 4
Description: as for outcome 7
Time Frame: Baseline (Day 1 Pre-dose), Week 2 and 4
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
micromol/L
  Week 2: number analyzed (Participants) | 18 | 14 | 17 | 17
  Week 2 | 0.4 (3.71) | -1.1 (1.70) | -1.3 (2.97) | 0.4 (4.14)
  Week 4: number analyzed (Participants) | 15 | 12 | 17 | 17
  Week 4 | 0.6 (2.82) | -1.7 (3.31) | -0.4 (3.33) | -0.4 (6.10)

12. Secondary Outcome: Change From Baseline in High Sensitivity C-reactive Protein (hsCRP) at Week 2 and Week 4
Description: as for outcome 7
Time Frame: Baseline (Day 1 Pre-dose), Week 2 and 4
Population: ITT population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: miligram per litre (mg/L)
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
miligram per litre (mg/L)
  Week 2: number analyzed (Participants) | 18 | 13 | 17 | 18
  Week 2 | 6.13 (32.236) | 2.35 (6.973) | -1.00 (13.878) | 4.32 (12.337)
  Week 4: number analyzed (Participants) | 15 | 11 | 16 | 17
  Week 4 | 0.21 (2.212) | 0.65 (3.383) | -2.09 (11.708) | 1.76 (9.378)

13. Secondary Outcome: Change From Baseline in Hematocrit and Reticulocytes Over 4 Weeks
Description: as for outcome 7
Time Frame: Baseline (Day 1 pre-dose), Week 1, 2, 3, and 4
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
Ratio
  Hematocrit, Week 1: number analyzed (Participants) | 19 | 16 | 18 | 17
  Hematocrit, Week 1 | -0.15 (1.385) | -0.29 (1.976) | -0.35 (0.941) | 0.39 (1.616)
  Hematocrit, Week 2: number analyzed (Participants) | 17 | 13 | 16 | 18
  Hematocrit, Week 2 | 0.35 (1.854) | 0.11 (1.570) | 0.24 (1.683) | 1.64 (2.103)
  Hematocrit, Week 3: number analyzed (Participants) | 18 | 12 | 17 | 17
  Hematocrit, Week 3 | -0.24 (1.752) | -0.56 (1.148) | 0.08 (1.406) | 2.11 (2.257)
  Hematocrit, Week 4: number analyzed (Participants) | 15 | 11 | 16 | 16
  Hematocrit, Week 4 | -0.50 (1.958) | -0.14 (1.204) | 1.16 (2.566) | 3.38 (2.052)
  Reticulocyte, Week 1: number analyzed (Participants) | 19 | 16 | 18 | 17
  Reticulocyte, Week 1 | 0.05 (0.494) | 0.24 (0.443) | 0.46 (0.725) | 0.95 (0.626)
  Reticulocyte, Week 2: number analyzed (Participants) | 17 | 13 | 16 | 18
  Reticulocyte, Week 2 | 0.01 (0.474) | 0.32 (0.458) | 0.12 (0.685) | 0.85 (0.633)
  Reticulocyte, Week 3: number analyzed (Participants) | 18 | 12 | 17 | 17
  Reticulocyte, Week 3 | 0.13 (0.479) | 0.23 (0.308) | 0.15 (0.634) | 0.45 (0.525)
  Reticulocyte, Week 4: number analyzed (Participants) | 15 | 11 | 16 | 16
  Reticulocyte, Week 4 | -0.07 (0.390) | 0.11 (0.375) | -0.07 (0.660) | 0.49 (0.532)

14. Secondary Outcome: Change From Baseline in Erythropoietin at Week 2 and Week 4
Description: Blood samples for erythropoietin were collected at Day 1 (pre-dose), Week 2 (first samples was collected approximately between 4 to 8 h and then 1 and 3 h after this fist sample) and Week 4 (Pre-dose and 3 h post-dose). The change from Baseline was calculated by subtracting the Baseline value from the individual post-dose visit values.
Time Frame: Baseline (Day 1 Pre-dose), Week 2 and 4
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per litre (U/L)
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
Units per litre (U/L)
  Week 2, 4-8 Hours Post-Dose: number analyzed (Participants) | 17 | 13 | 16 | 18
  Week 2, 4-8 Hours Post-Dose | 0.721 (6.1773) | 1.022 (4.4319) | 3.622 (10.0551) | 13.267 (17.8580)
  Week 2, 5-9 Hours, Post Dose: number analyzed (Participants) | 16 | 13 | 16 | 18
  Week 2, 5-9 Hours, Post Dose | 1.541 (6.6890) | 1.027 (4.3872) | 4.612 (10.9494) | 15.800 (18.5065)
  Week 2, 7-11 Hours, Post Dose: number analyzed (Participants) | 15 | 12 | 16 | 18
  Week 2, 7-11 Hours, Post Dose | 0.437 (5.4935) | 0.538 (4.5382) | 6.630 (13.4120) | 20.100 (18.5656)
  Week 4, Pre-dose: number analyzed (Participants) | 15 | 10 | 15 | 16
  Week 4, Pre-dose | 6.644 (17.6483) | 0.014 (3.9986) | 0.814 (6.8894) | 2.975 (7.5732)
  Week 4, 3 Hour Post-Dose: number analyzed (Participants) | 15 | 9 | 15 | 16
  Week 4, 3 Hour Post-Dose | 6.346 (18.2978) | 1.039 (5.1686) | -0.075 (7.6779) | 2.102 (6.9180)

15. Secondary Outcome: Change From Baseline in Red Blood Cells Count Over 4 Weeks
Description: as for outcome 7
Time Frame: Baseline (Day 1 pre-dose), week 1, 2, 3, 4
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells /L
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
10^12 cells /L
  Week 1: number analyzed (Participants) | 19 | 16 | 18 | 17
  Week 1 | -0.01 (0.137) | -0.03 (0.181) | -0.03 (0.113) | 0.04 (0.162)
  Week 2: number analyzed (Participants) | 17 | 13 | 16 | 18
  Week 2 | 0.02 (0.181) | 0.03 (0.160) | 0.01 (0.165) | 0.14 (0.225)
  Week 3: number analyzed (Participants) | 18 | 12 | 17 | 17
  Week 3 | -0.03 (0.193) | -0.02 (0.136) | -0.02 (0.147) | 0.16 (0.223)
  Week 4: number analyzed (Participants) | 15 | 11 | 16 | 16
  Week 4 | -0.05 (0.181) | 0.01 (0.145) | 0.09 (0.254) | 0.33 (0.209)

16. Secondary Outcome: Change From Baseline in Vascular Endothelial Growth Factor (VEGF) at Week 2 and Week 4
Description: Blood samples for VEGF were collected at Day 1 (pre-dose), Week 2 (first samples was collected approximately between 4 to 8 h and then 1 and 3 h after this fist sample) and Week 4 (Pre-dose and 3 h post-dose). Baseline was the Day 1 pre-dose value. The change from baseline was calculated by subtracting the baseline value from the individual post-dose visit values.
Time Frame: Baseline (Pre-dose), week 2 and 4
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram per litre (ng/L)
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 19 | 16 | 18 | 18
Nanogram per litre (ng/L)
  WEEK 2, 4-8 HOURS POST-DOSE: number analyzed (Participants) | 17 | 13 | 16 | 18
  WEEK 2, 4-8 HOURS POST-DOSE | -12.09 (62.267) | -17.23 (56.519) | -19.55 (88.167) | 20.38 (60.840)
  WEEK 2, 5-9 HOURS, POST DOSE: number analyzed (Participants) | 16 | 13 | 16 | 18
  WEEK 2, 5-9 HOURS, POST DOSE | -23.04 (104.309) | -18.21 (33.258) | -11.80 (100.745) | 8.38 (39.975)
  WEEK 2, 7-11 HOURS, POST DOSE: number analyzed (Participants) | 15 | 12 | 15 | 18
  WEEK 2, 7-11 HOURS, POST DOSE | -41.40 (133.098) | -30.56 (58.602) | -17.88 (89.793) | 14.40 (41.786)
  WEEK 4, PRE-DOSE: number analyzed (Participants) | 15 | 10 | 15 | 14
  WEEK 4, PRE-DOSE | -39.69 (114.265) | 65.89 (161.068) | -7.47 (29.058) | -1.48 (30.874)
  WEEK 4, 3 HOUR POST-DOSE: number analyzed (Participants) | 15 | 9 | 15 | 15
  WEEK 4, 3 HOUR POST-DOSE | -43.33 (136.048) | 0.77 (37.861) | -3.87 (36.521) | 5.56 (41.400)

17. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE was defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE include AEs those result in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Up to 6 weeks
Population: The Safety Population comprised of all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
Participants
  Any AEs | 9 | 10 | 5 | 6
  Any SAEs | 1 | 0 | 2 | 1

18. Secondary Outcome: Number of Participants Discontinuing the Study Treatment Due to AEs
Description: AE was defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE include AEs those result in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. number of participants discontinuing the study treatment due to AEs.
Time Frame: Up to 6 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
Participants | 1 | 1 | 0 | 0

19. Secondary Outcome: Absolute Values of Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST), Creatine Kinase (CK) at Baseline (Day 1), Week 2, 4, and 6
Description: Clinical chemistry parameters including ALT, ALP, AST, CK were assessed at Baseline (Day 1 pre-dose), Week 2, 4, and at follow-up visit (Week 6).
Time Frame: Baseline (Day 1 pre-dose), Week 2, 4, and 6
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International Units per litre (IU/L)
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
International Units per litre (IU/L)
  ALT, Day 1: number analyzed (Participants) | 18 | 17 | 17 | 19
  ALT, Day 1 | 11.8 (4.85) | 13.8 (5.74) | 18.8 (14.40) | 16.2 (7.08)
  ALT, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  ALT, Week 2 | 10.8 (3.68) | 12.4 (5.28) | 20.1 (23.79) | 14.1 (6.26)
  ALT, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  ALT, Week 4 | 11.4 (3.61) | 14.6 (8.92) | 22.2 (31.12) | 13.2 (4.25)
  ALT, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  ALT, Week 6 | 10.1 (3.11) | 14.9 (8.57) | 16.9 (9.55) | 16.5 (6.16)
  ALP, Day 1: number analyzed (Participants) | 18 | 17 | 17 | 19
  ALP, Day 1 | 86.6 (28.50) | 95.6 (31.47) | 97.7 (30.48) | 85.9 (31.47)
  ALP, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  ALP, Week 2 | 84.3 (23.73) | 91.5 (28.90) | 92.2 (24.56) | 87.2 (31.54)
  ALP, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  ALP, Week 4 | 84.1 (23.02) | 90.4 (30.57) | 92.6 (23.51) | 90.1 (34.71)
  ALP, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  ALP, Week 6 | 83.9 (21.32) | 89.2 (31.38) | 87.1 (20.13) | 92.4 (37.56)
  AST, Day 1: number analyzed (Participants) | 18 | 17 | 17 | 19
  AST, Day 1 | 16.7 (4.51) | 19.1 (5.00) | 22.9 (14.70) | 18.7 (6.68)
  AST, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  AST, Week 2 | 16.1 (3.21) | 17.5 (5.42) | 26.1 (22.66) | 19.0 (7.08)
  AST, Week 4: number analyzed (Participants) | 14 | 13 | 16 | 17
  AST, Week 4 | 15.6 (2.44) | 18.2 (5.37) | 26.7 (29.90) | 17.4 (6.06)
  AST, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  AST, Week 6 | 15.2 (2.81) | 20.1 (5.69) | 21.4 (7.12) | 19.8 (6.77)
  CK, Day 1: number analyzed (Participants) | 18 | 17 | 17 | 19
  CK, Day 1 | 101.6 (73.24) | 132.4 (127.75) | 159.4 (129.56) | 94.4 (55.38)
  CK, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  CK, Week 2 | 86.7 (51.04) | 130.8 (124.04) | 150.2 (92.89) | 100.0 (78.25)
  CK, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  CK, Week 4 | 94.4 (53.19) | 114.2 (81.35) | 136.4 (111.22) | 83.1 (78.25)
  CK, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  CK, Week 6 | 90.6 (60.11) | 132.2 (97.34) | 137.4 (82.22) | 130.9 (269.29)

20. Secondary Outcome: Absolute Values of Albumin, Apolipoprotein A1, Apolipoprotein Total, Total Protein at Baseline (Day 1), Week 2, 4, and 6
Description: Clinical chemistry parameters including albumin, apolipoprotein A1, apolipoprotein total, total protein were assessed at Baseline (Day 1 pre-dose), Week 2, 4, and at follow-up visit (Week 6).
Time Frame: Baseline (Day 1 pre-dose), Week 2, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
G/L
  Albumin, Day 1: number analyzed (Participants) | 18 | 17 | 17 | 19
  Albumin, Day 1 | 39.8 (3.37) | 40.9 (4.12) | 39.7 (4.38) | 39.8 (3.50)
  Albumin, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Albumin, Week 2 | 40.8 (3.91) | 40.3 (5.31) | 38.8 (4.38) | 40.1 (3.54)
  Albumin, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Albumin, Week 4 | 40.6 (3.00) | 41.3 (3.68) | 39.1 (4.33) | 39.2 (4.10)
  Albumin, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Albumin, Week 6 | 40.0 (4.21) | 39.9 (5.04) | 40.6 (3.22) | 38.9 (3.33)
  Apolipoprotein A1, Day 1: number analyzed (Participants) | 18 | 17 | 16 | 19
  Apolipoprotein A1, Day 1 | 1.481 (0.2352) | 1.515 (0.2546) | 1.461 (0.3561) | 1.572 (0.4178)
  Apolipoprotein A1, Week 2: number analyzed (Participants) | 17 | 15 | 18 | 18
  Apolipoprotein A1, Week 2 | 1.418 (0.1732) | 1.472 (0.2901) | 1.469 (0.3142) | 1.370 (0.3831)
  Apolipoprotein A1, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Apolipoprotein A1, Week 4 | 1.482 (0.1712) | 1.452 (0.3034) | 1.436 (0.2553) | 1.405 (0.4564)
  Apolipoprotein A1, Week 6: number analyzed (Participants) | 15 | 15 | 16 | 17
  Apolipoprotein A1, Week 6 | 1.472 (0.1921) | 1.501 (0.2482) | 1.468 (0.2514) | 1.492 (0.4378)
  Apolipoprotein Total, Day 1: number analyzed (Participants) | 18 | 17 | 16 | 19
  Apolipoprotein Total, Day 1 | 0.794 (0.2278) | 0.936 (0.2645) | 0.788 (0.2419) | 0.792 (0.2884)
  Apolipoprotein Total, Week 2: number analyzed (Participants) | 17 | 15 | 18 | 18
  Apolipoprotein Total, Week 2 | 0.754 (0.2190) | 0.901 (0.2529) | 0.733 (0.1921) | 0.751 (0.3278)
  Apolipoprotein Total, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Apolipoprotein Total, Week 4 | 0.720 (0.1727) | 0.888 (0.2535) | 0.724 (0.2071) | 0.743 (0.2921)
  Apolipoprotein Total, Week 6: number analyzed (Participants) | 15 | 15 | 16 | 17
  Apolipoprotein Total, Week 6 | 0.732 (0.1843) | 0.872 (0.2062) | 0.757 (0.2286) | 0.776 (0.3036)
  Total Protein, Day 1: number analyzed (Participants) | 18 | 17 | 17 | 19
  Total Protein, Day 1 | 69.4 (8.53) | 71.1 (6.41) | 68.5 (5.50) | 67.7 (4.90)
  Total Protein, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Total Protein, Week 2 | 70.8 (9.24) | 70.1 (7.81) | 66.4 (4.26) | 68.3 (4.54)
  Total Protein, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Total Protein, Week 4 | 70.7 (10.87) | 71.8 (6.53) | 66.9 (4.24) | 67.6 (6.77)
  Total Protein, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Total Protein, Week 6 | 69.8 (9.83) | 69.7 (8.36) | 68.3 (3.26) | 66.9 (4.88)

21. Secondary Outcome: Absolute Values of Calcium, Chloride, Cholesterol, Glucose, Inorganic Phosphorus, Potassium, Sodium at Baseline (Day 1), Week 2, 4, and 6
Description: Clinical chemistry parameters including calcium, chloride, cholesterol, glucose, inorganic phosphorus, potassium, sodium were assessed at Baseline (Day 1 pre-dose), Week 2, 4, and at follow-up visit (Week 6).
Time Frame: Baseline (Day 1 pre-dose), Week 2, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimol per Litre (MMOL/L)
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
Millimol per Litre (MMOL/L)
  Calcium, Day 1: number analyzed (Participants) | 18 | 17 | 17 | 19
  Calcium, Day 1 | 2.258 (0.1026) | 2.296 (0.1404) | 2.259 (0.1537) | 2.335 (0.1351)
  Calcium, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Calcium, Week 2 | 2.299 (0.0915) | 2.298 (0.1472) | 2.331 (0.1293) | 2.347 (0.1510)
  Calcium, Week 4: number analyzed (Participants) | 14 | 13 | 16 | 16
  Calcium, Week 4 | 2.274 (0.0872) | 2.302 (0.1234) | 2.301 (0.0922) | 2.348 (0.1610)
  Calcium, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Calcium, Week 6 | 2.255 (0.1049) | 2.331 (0.1861) | 2.309 (0.1489) | 2.322 (0.1360)
  Chloride, Day 1: number analyzed (Participants) | 18 | 17 | 17 | 19
  Chloride, Day 1 | 105.4 (3.05) | 103.1 (3.83) | 103.9 (5.98) | 104.7 (5.11)
  Chloride, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Chloride, Week 2 | 105.6 (2.69) | 104.2 (4.31) | 103.6 (6.31) | 103.1 (5.90)
  Chloride, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Chloride, Week 4 | 106.6 (3.91) | 105.0 (4.43) | 104.0 (5.56) | 106.4 (3.97)
  Chloride, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Chloride, Week 6 | 106.7 (3.52) | 105.3 (3.99) | 103.8 (6.19) | 104.2 (3.90)
  Cholesterol, Day 1: number analyzed (Participants) | 18 | 17 | 17 | 19
  Cholesterol, Day 1 | 4.147 (0.9085) | 4.632 (1.2160) | 4.088 (1.1424) | 4.411 (1.4333)
  Cholesterol, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Cholesterol, Week 2 | 3.997 (0.7547) | 4.623 (1.1469) | 3.800 (0.8787) | 4.282 (1.5566)
  Cholesterol, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Cholesterol, Week 4 | 3.893 (0.5880) | 4.448 (1.0808) | 3.776 (0.9276) | 4.091 (1.4236)
  Cholesterol, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Cholesterol, Week 6 | 3.944 (0.6613) | 4.520 (1.0775) | 3.928 (1.0253) | 4.406 (1.4561)
  Glucose, Day 1: number analyzed (Participants) | 18 | 17 | 17 | 19
  Glucose, Day 1 | 6.97 (3.082) | 9.11 (5.189) | 9.46 (4.840) | 7.75 (3.077)
  Glucose, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Glucose, Week 2 | 6.78 (3.333) | 8.48 (4.322) | 9.64 (4.160) | 9.42 (6.596)
  Glucose, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Glucose, Week 4 | 6.49 (3.246) | 9.03 (4.940) | 8.63 (2.653) | 6.71 (2.162)
  Glucose, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Glucose, Week 6 | 8.88 (5.534) | 8.34 (3.503) | 9.14 (4.243) | 7.81 (3.506)
  Phosphorus, inorganic, Day 1: number analyzed (Participants) | 18 | 17 | 17 | 19
  Phosphorus, inorganic, Day 1 | 1.325 (0.2686) | 1.364 (0.2545) | 1.403 (0.3165) | 1.313 (0.2655)
  Phosphorus, inorganic, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Phosphorus, inorganic, Week 2 | 1.309 (0.2116) | 1.421 (0.2848) | 1.435 (0.3297) | 1.285 (0.2871)
  Phosphorus, inorganic, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Phosphorus, inorganic, Week 4 | 1.293 (0.2235) | 1.388 (0.2922) | 1.403 (0.2660) | 1.244 (0.2674)
  Phosphorus, inorganic, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Phosphorus, inorganic, Week 6 | 1.319 (0.2810) | 1.345 (0.2527) | 1.366 (0.3567) | 1.203 (0.2322)
  Potassium, Day 1: number analyzed (Participants) | 18 | 17 | 17 | 19
  Potassium, Day 1 | 4.57 (0.452) | 4.65 (0.632) | 4.65 (0.489) | 4.63 (0.498)
  Potassium, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Potassium, Week 2 | 4.67 (0.410) | 4.61 (0.703) | 4.71 (0.627) | 4.62 (0.593)
  Potassium, Week 4: number analyzed (Participants) | 14 | 13 | 16 | 17
  Potassium, Week 4 | 4.54 (0.460) | 4.61 (0.468) | 4.56 (0.671) | 4.42 (0.602)
  Potassium, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Potassium, Week 6 | 4.56 (0.510) | 4.58 (0.496) | 4.70 (0.520) | 4.65 (0.624)
  Sodium, Day 1: number analyzed (Participants) | 18 | 17 | 17 | 19
  Sodium, Day 1 | 140.1 (2.65) | 137.8 (3.00) | 137.5 (3.92) | 138.6 (3.45)
  Sodium, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Sodium, Week 2 | 139.8 (2.60) | 137.9 (2.00) | 138.2 (3.88) | 137.5 (4.62)
  Sodium, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Sodium, Week 4 | 140.6 (3.13) | 139.2 (2.65) | 138.5 (3.59) | 140.2 (3.53)
  Sodium, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Sodium, Week 6 | 140.3 (2.46) | 139.4 (2.13) | 137.9 (4.65) | 138.8 (2.83)

22. Secondary Outcome: Absolute Values of Creatinine, Direct Bilirubin, Indirect Bilirubin, Total Bilirubin at Baseline (Day 1), Week 2, 4, and 6
Description: Clinical chemistry parameters including creatinine, direct bilirubin, indirect bilirubin, total bilirubin were assessed at Baseline (Day 1 pre-dose), Week 2, 4, and at follow-up visit (Week 6).
Time Frame: Baseline (Day 1 pre-dose), Week 2, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromol/L
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
Micromol/L
  Creatinine, Day 1: number analyzed (Participants) | 18 | 17 | 17 | 19
  Creatinine, Day 1 | 250.67 (110.117) | 237.05 (91.762) | 274.34 (146.092) | 237.43 (128.461)
  Creatinine, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Creatinine, Week 2 | 235.92 (86.636) | 245.16 (91.810) | 267.07 (166.480) | 217.84 (112.543)
  Creatinine, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Creatinine, Week 4 | 242.21 (106.796) | 250.10 (101.583) | 254.86 (149.148) | 209.76 (109.374)
  Creatinine, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Creatinine, Week 6 | 244.43 (94.682) | 238.07 (99.771) | 254.86 (171.772) | 219.50 (111.645)
  Direct bilirubin, Day 1: number analyzed (Participants) | 17 | 17 | 17 | 19
  Direct bilirubin, Day 1 | 1.9 (1.11) | 2.1 (1.50) | 2.1 (1.11) | 1.6 (1.07)
  Direct bilirubin, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Direct bilirubin, Week 2 | 1.5 (1.12) | 1.7 (1.50) | 1.8 (0.66) | 2.1 (1.11)
  Direct bilirubin, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Direct bilirubin, Week 4 | 1.6 (0.85) | 1.8 (1.54) | 1.9 (0.86) | 1.9 (1.11)
  Direct bilirubin, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Direct bilirubin, Week 6 | 1.8 (1.44) | 1.8 (1.61) | 1.8 (0.68) | 2.1 (0.86)
  Indirect bilirubin, Day 1: number analyzed (Participants) | 17 | 17 | 17 | 19
  Indirect bilirubin, Day 1 | 4.0 (1.41) | 4.4 (1.46) | 4.4 (1.46) | 4.6 (1.34)
  Indirect bilirubin, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Indirect bilirubin, Week 2 | 5.1 (2.01) | 4.5 (1.55) | 4.8 (1.74) | 4.6 (2.09)
  Indirect bilirubin, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Indirect bilirubin, Week 4 | 4.3 (1.07) | 4.2 (1.30) | 4.8 (1.74) | 4.9 (1.75)
  Indirect bilirubin, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Indirect bilirubin, Week 6 | 4.4 (1.67) | 5.0 (2.42) | 4.8 (1.24) | 3.8 (0.97)
  Total bilirubin, Day 1: number analyzed (Participants) | 17 | 17 | 17 | 19
  Total bilirubin, Day 1 | 5.9 (1.50) | 6.5 (0.87) | 6.5 (1.94) | 6.2 (1.62)
  Total bilirubin, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Total bilirubin, Week 2 | 6.6 (2.09) | 6.1 (1.41) | 6.6 (1.97) | 6.7 (2.34)
  Total bilirubin, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Total bilirubin, Week 4 | 5.9 (1.23) | 6.0 (1.15) | 6.7 (1.99) | 6.8 (2.35)
  Total bilirubin, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Total bilirubin, Week 6 | 6.1 (1.36) | 6.8 (3.19) | 6.5 (1.37) | 5.9 (1.50)

23. Secondary Outcome: Absolute Values of Urine Total Protein/Creatinine Ratio at Baseline (Day 1), Week 2, 4, and 6
Description: Absolute values of urine total protein/creatinine ratio at Baseline (Day 1), Week 2, 4, and follow-up (week 6) were reported.
Time Frame: Baseline (Day 1), Week 2, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mg/MMOL
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
mg/MMOL
  Urine Total Protein/Creatinine ratio, Day 1: number analyzed (Participants) | 14 | 14 | 13 | 16
  Urine Total Protein/Creatinine ratio, Day 1 | 226.00 (268.727) | 205.73 (366.100) | 342.39 (518.396) | 211.58 (241.306)
  Urine Total Protein/Creatinine ratio, Week 2: number analyzed (Participants) | 15 | 14 | 15 | 13
  Urine Total Protein/Creatinine ratio, Week 2 | 170.41 (194.898) | 207.82 (281.943) | 194.14 (314.152) | 149.08 (135.788)
  Urine Total Protein/Creatinine ratio, Week 4: number analyzed (Participants) | 14 | 13 | 16 | 15
  Urine Total Protein/Creatinine ratio, Week 4 | 114.71 (130.867) | 169.31 (262.401) | 196.37 (326.453) | 219.47 (280.924)
  Urine Total Protein/Creatinine ratio, Week 6: number analyzed (Participants) | 14 | 12 | 13 | 13
  Urine Total Protein/Creatinine ratio, Week 6 | 232.80 (381.556) | 162.81 (275.606) | 175.16 (314.341) | 160.01 (192.595)

24. Secondary Outcome: Change From Baseline Values of ALT, ALP, AST, CK at Week 2, 4, and 6
Description: Baseline values were recorded on Day 1. If the Day 1 value was missing, the last non-missing value from week -1 or week-2 was represented as the Baseline value. The change from Baseline was calculated by subtracting the Baseline value from the individual post-dose visit values. Change from Baseline values of ALT, AST, ALP and CK at Week 2, 4, and 6
Time Frame: Baseline (Day 1), Week 2, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
IU/L
  ALT, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  ALT, Week 2 | -1.1 (2.89) | -1.2 (3.32) | 3.9 (21.85) | -1.9 (4.16)
  ALT, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  ALT, Week 4 | 0.1 (3.38) | 0.7 (6.79) | 6.0 (29.33) | -2.8 (7.68)
  ALT, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  ALT, Week 6 | -1.3 (3.09) | 0.7 (4.19) | 0.4 (7.51) | 0.5 (9.02)
  ALP, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  ALP, Week 2 | 0.8 (10.25) | -2.8 (12.11) | -1.2 (12.31) | 2.7 (10.52)
  ALP, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  ALP, Week 4 | 1.1 (8.92) | -4.8 (10.49) | -0.8 (18.42) | 2.6 (8.15)
  ALP, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  ALP, Week 6 | -1.9 (11.51) | -6.4 (14.19) | -5.7 (19.41) | 4.9 (13.40)
  AST, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  AST, Week 2 | -0.9 (2.66) | -1.7 (3.51) | 4.7 (21.33) | 0.1 (3.92)
  AST, Week 4: number analyzed (Participants) | 14 | 13 | 16 | 17
  AST, Week 4 | -1.3 (3.24) | -0.5 (4.37) | 5.1 (28.99) | -1.1 (4.70)
  AST, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  AST, Week 6 | -1.6 (3.03) | -0.1 (5.92) | -0.3 (7.89) | 1.4 (4.66)
  CK, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  CK, Week 2 | -18.7 (34.45) | 7.9 (137.74) | 1.2 (61.44) | 4.4 (53.00)
  CK, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  CK, Week 4 | -21.4 (57.79) | -8.5 (90.90) | -12.6 (66.40) | -7.5 (39.31)
  CK, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  CK, Week 6 | -19.1 (37.64) | -9.4 (97.00) | -5.1 (63.93) | 40.4 (240.54)

25. Secondary Outcome: Change From Baseline Values of Albumin, Apolipoprotein A1, Apolipoprotein Total, Total Protein at Week 2, 4, and 6
Description: Baseline values were recorded on Day 1 (Pre dose). If the Day 1 value was missing, the last non-missing value from week -1 or week-2 was represented as the baseline value. The change from baseline was calculated by subtracting the baseline value from the individual post-dose visit values. Change from Baseline values of albumin, apolipoprotein A1, apolipoprotein total, total protein at Week 2, 4, and 6 were reported.
Time Frame: Baseline (Day 1), Week 2, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
G/L
  Albumin, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Albumin, Week 2 | 0.7 (1.86) | -0.5 (1.92) | -0.9 (2.12) | -0.4 (2.12)
  Albumin, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Albumin, Week 4 | 0.4 (2.03) | -0.2 (2.08) | -0.6 (0.87) | -0.6 (2.71)
  Albumin, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Albumin, Week 6 | 0.2 (2.01) | -1.2 (2.08) | 0.1 (1.89) | -1.0 (2.65)
  Apolipoprotein A1, Week 2: number analyzed (Participants) | 17 | 15 | 16 | 18
  Apolipoprotein A1, Week 2 | -0.045 (0.0887) | -0.063 (0.1386) | -0.023 (0.1754) | -0.197 (0.1641)
  Apolipoprotein A1, Week 4: number analyzed (Participants) | 14 | 13 | 15 | 17
  Apolipoprotein A1, Week 4 | -0.011 (0.1144) | -0.061 (0.1198) | -0.025 (0.1932) | -0.163 (0.2133)
  Apolipoprotein A1, Week 6: number analyzed (Participants) | 15 | 15 | 14 | 17
  Apolipoprotein A1, Week 6 | -0.009 (0.1287) | -0.026 (0.1408) | -0.011 (0.1618) | -0.076 (0.2743)
  Apolipoprotein total, Week 2: number analyzed (Participants) | 17 | 15 | 16 | 18
  Apolipoprotein total, Week 2 | -0.016 (0.0775) | -0.067 (0.1254) | -0.051 (0.1312) | -0.048 (0.1488)
  Apolipoprotein total, Week 4: number analyzed (Participants) | 14 | 13 | 15 | 17
  Apolipoprotein total, Week 4 | -0.036 (0.0954) | -0.051 (0.0910) | -0.055 (0.1852) | -0.024 (0.2123)
  Apolipoprotein total, Week 6: number analyzed (Participants) | 15 | 15 | 14 | 17
  Apolipoprotein total, Week 6 | -0.007 (0.0952) | -0.077 (0.1685) | 0.014 (0.2147) | 0.009 (0.2194)
  Total protein, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Total protein, Week 2 | 1.1 (3.04) | -0.7 (3.03) | -1.3 (3.64) | -0.2 (2.79)
  Total protein, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Total protein, Week 4 | 0.5 (3.18) | -0.1 (3.64) | -0.8 (2.65) | 0.2 (4.50)
  Total protein, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Total protein, Week 6 | 0.4 (2.73) | -1.5 (3.20) | -0.3 (2.44) | -0.6 (2.92)

26. Secondary Outcome: Change From Baseline Values of Calcium, Chloride, Cholesterol, Glucose, Inorganic Phosphorus, Potassium, Sodium at Week 2, 4, and 6
Description: Baseline values were recorded on Day 1. If the Day 1 value was missing, the last non-missing value from week -1 or week-2 was represented as the baseline value. The change from baseline was calculated by subtracting the baseline value from the individual post-dose visit values. Change from Baseline values of calcium, chloride, cholesterol, glucose, inorganic phosphorus, potassium, sodium at Week 2, 4, and 6 were reported.
Time Frame: Baseline (Day 1), Week 2, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: MMOL/L
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
MMOL/L
  Calcium, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Calcium, Week 2 | 0.044 (0.0686) | 0.017 (0.0767) | 0.032 (0.0977) | 0.014 (0.0717)
  Calcium, Week 4: number analyzed (Participants) | 14 | 13 | 16 | 16
  Calcium, Week 4 | 0.021 (0.1088) | 0.008 (0.0870) | -0.000 (0.0641) | 0.010 (0.0719)
  Calcium, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Calcium, Week 6 | 0.000 (0.1073) | 0.019 (0.1192) | -0.001 (0.0959) | -0.014 (0.0514)
  Chloride, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Chloride, Week 2 | 0.0 (3.59) | 0.9 (3.34) | -0.5 (4.95) | -1.5 (3.54)
  Chloride, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Chloride, Week 4 | 1.4 (2.84) | 1.8 (3.26) | -0.1 (3.43) | 0.9 (3.69)
  Chloride, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Chloride, Week 6 | 1.1 (2.95) | 1.9 (3.51) | -0.1 (3.94) | -1.3 (3.37)
  Cholesterol, Week 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cholesterol, Week 1 | 0.050 (NA) — Only one participant was analyzed. Dispersion could not be calculated. |  |  |
  Cholesterol, Week 2: number analyzed (Participants) | 17 | 15 | 16 | 17
  Cholesterol, Week 2 | -0.029 (0.2948) | -0.150 (0.5398) | -0.256 (0.3907) | -0.244 (0.6290)
  Cholesterol, Week 4: number analyzed (Participants) | 14 | 13 | 16 | 17
  Cholesterol, Week 4 | -0.136 (0.3060) | -0.195 (0.4310) | -0.288 (0.6412) | -0.285 (0.8511)
  Cholesterol, Week 6: number analyzed (Participants) | 16 | 15 | 15 | 17
  Cholesterol, Week 6 | -0.134 (0.4704) | -0.223 (0.7452) | -0.040 (0.8412) | 0.029 (0.7814)
  Glucose, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Glucose, Week 2 | 0.35 (3.025) | -0.59 (5.940) | 0.13 (4.375) | 1.67 (5.073)
  Glucose, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Glucose, Week 4 | 0.01 (2.893) | -0.21 (3.809) | -0.88 (3.968) | -0.51 (1.957)
  Glucose, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Glucose, Week 6 | 1.89 (3.913) | 0.53 (3.725) | -0.57 (5.339) | 0.59 (2.585)
  Inorganic phosphorus, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Inorganic phosphorus, Week 2 | 0.012 (0.1420) | 0.065 (0.1536) | 0.032 (0.2277) | 0.026 (0.2122)
  Inorganic phosphorus, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Inorganic phosphorus, Week 4 | 0.025 (0.1718) | 0.015 (0.1784) | 0.000 (0.2430) | -0.032 (0.1828)
  Inorganic phosphorus, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Inorganic phosphorus, Week 6 | 0.003 (0.3041) | -0.031 (0.1345) | -0.009 (0.2478) | -0.074 (0.1161)
  Potassium, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Potassium, Week 2 | 0.10 (0.420) | 0.01 (0.500) | 0.08 (0.558) | -0.02 (0.437)
  Potassium, Week 4: number analyzed (Participants) | 14 | 13 | 16 | 17
  Potassium, Week 4 | 0.05 (0.470) | -0.02 (0.559) | -0.04 (0.488) | -0.23 (0.541)
  Potassium, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Potassium, Week 6 | 0.05 (0.601) | -0.05 (0.385) | 0.06 (0.346) | 0.01 (0.439)
  Sodium, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Sodium, Week 2 | -0.3 (2.42) | 0.1 (2.53) | 0.3 (2.80) | -0.9 (2.86)
  Sodium, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Sodium, Week 4 | 0.5 (3.78) | 1.6 (2.84) | 0.6 (2.96) | 1.3 (3.72)
  Sodium, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Sodium, Week 6 | -0.2 (2.29) | 1.3 (2.87) | 0.1 (3.04) | -0.1 (2.83)

27. Secondary Outcome: Change From Baseline Values of Creatinine, Direct Bilirubin, Indirect Bilirubin, Total Bilirubin at Week 2, 4, and 6
Description: Baseline values were recorded on Day 1. If the Day 1 value was missing, the last non-missing value from week -1 or week-2 was represented as the baseline value. The change from baseline was calculated by subtracting the baseline value from the individual post-dose visit values. Change from Baseline values of creatinine, direct bilirubin, indirect bilirubin, total bilirubin at Week 2, 4, and 6 were reported.
Time Frame: Baseline (Day 1), Week 2, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromol/L
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
Micromol/L
  Creatinine, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Creatinine, Week 2 | -1.41 (22.366) | -0.99 (29.854) | 10.78 (51.170) | -2.60 (18.802)
  Creatinine, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Creatinine, Week 4 | 11.79 (20.853) | 1.65 (18.800) | -1.44 (37.000) | -16.96 (23.293)
  Creatinine, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Creatinine, Week 6 | 0.71 (46.295) | -5.01 (41.477) | 7.24 (58.581) | -7.23 (29.816)
  Direct bilirubin, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Direct bilirubin, Week 2 | -0.5 (1.66) | -0.3 (1.99) | -0.4 (1.06) | 0.4 (1.27)
  Direct bilirubin, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Direct bilirubin, Week 4 | -0.6 (1.65) | -0.2 (1.74) | -0.2 (0.97) | 0.2 (1.20)
  Direct bilirubin, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Direct bilirubin, Week 6 | -0.4 (1.67) | -0.5 (1.13) | -0.4 (1.31) | 0.5 (0.87)
  Indirect bilirubin, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Indirect bilirubin, Week 2 | 1.2 (2.13) | 0.1 (2.40) | 0.5 (1.33) | -0.1 (2.39)
  Indirect bilirubin, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Indirect bilirubin, Week 4 | 0.4 (1.60) | -0.2 (2.17) | 0.5 (1.66) | 0.5 (1.66)
  Indirect bilirubin, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Indirect bilirubin, Week 6 | 0.4 (2.09) | 0.9 (2.17) | 0.3 (1.61) | -0.7 (0.99)
  Total bilirubin, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 17
  Total bilirubin, Week 2 | 0.7 (1.72) | -0.3 (1.03) | 0.1 (1.32) | 0.2 (2.33)
  Total bilirubin, Week 4: number analyzed (Participants) | 14 | 13 | 17 | 17
  Total bilirubin, Week 4 | -0.1 (1.23) | -0.5 (0.88) | 0.2 (1.86) | 0.7 (1.21)
  Total bilirubin, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 17
  Total bilirubin, Week 6 | 0.0 (1.79) | 0.4 (2.53) | -0.1 (1.86) | -0.2 (0.66)

28. Secondary Outcome: Change From Baseline Values of Urine Total Protein/Creatinine Ratio at Week 2, 4, and 6
Description: Baseline values were recorded on Day 1. If the Day 1 value was missing, the last non-missing value from week -1 or week-2 was represented as the baseline value. The change from baseline was calculated by subtracting the baseline value from the individual post-dose visit values. Change from Baseline values of urine total protein/creatinine ratio at Week 2, 4, and 6 were reported.
Time Frame: Baseline (Day 1), Week 2, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: MG/MMOL
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
MG/MMOL
  Urine Total Protein/Creatinine ratio, Week 2: number analyzed (Participants) | 13 | 11 | 12 | 12
  Urine Total Protein/Creatinine ratio, Week 2 | 3.44 (39.792) | -38.83 (97.814) | -115.28 (265.028) | -77.98 (173.654)
  Urine Total Protein/Creatinine ratio, Week 4: number analyzed (Participants) | 10 | 10 | 12 | 13
  Urine Total Protein/Creatinine ratio, Week 4 | -20.56 (50.953) | 17.43 (58.837) | -99.40 (209.678) | 39.90 (86.729)
  Urine Total Protein/Creatinine ratio, Week 6: number analyzed (Participants) | 11 | 10 | 10 | 11
  Urine Total Protein/Creatinine ratio, Week 6 | 47.22 (185.115) | -26.73 (67.464) | -72.19 (187.792) | -41.40 (191.418)

29. Secondary Outcome: Absolute Values of Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count, WBC Count (Absolute) at Baseline, Week 1, 2, 3, 4, and 6
Description: Hematology parameters including Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet count, WBC count (absolute) were assessed at Baseline (Day 1 pre-dose), Week 2, 3, 4, and at follow-up visit (Week 6).
Time Frame: Baseline (Day 1 pre-dose), Week 1, 2, 3, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
10^9 cells/L
  Basophils, Day 1: number analyzed (Participants) | 18 | 17 | 16 | 18
  Basophils, Day 1 | 0.023 (0.0136) | 0.035 (0.0255) | 0.025 (0.0207) | 0.025 (0.0179)
  Basophils, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Basophils, Week 1 | 0.023 (0.0141) | 0.023 (0.0086) | 0.034 (0.0212) | 0.030 (0.0157)
  Basophils, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Basophils, Week 2 | 0.026 (0.0121) | 0.022 (0.0153) | 0.024 (0.0146) | 0.029 (0.0261)
  Basophils, Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  Basophils, Week 3 | 0.027 (0.0228) | 0.031 (0.0166) | 0.024 (0.0132) | 0.026 (0.0252)
  Basophils, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Basophils, Week 4 | 0.027 (0.0252) | 0.033 (0.0303) | 0.023 (0.0124) | 0.024 (0.0182)
  Basophils, Week 6: number analyzed (Participants) | 14 | 14 | 16 | 17
  Basophils, Week 6 | 0.024 (0.0122) | 0.029 (0.0138) | 0.023 (0.0134) | 0.024 (0.0141)
  Eosinophils, Day 1: number analyzed (Participants) | 18 | 17 | 16 | 18
  Eosinophils, Day 1 | 0.226 (0.2505) | 0.205 (0.0859) | 0.165 (0.1067) | 0.141 (0.0657)
  Eosinophils, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Eosinophils, Week 1 | 0.212 (0.2288) | 0.189 (0.1021) | 0.126 (0.1054) | 0.169 (0.0893)
  Eosinophils, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Eosinophils, Week 2 | 0.204 (0.2685) | 0.223 (0.1274) | 0.122 (0.0811) | 0.112 (0.0568)
  Eosinophils, Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  Eosinophils, Week 3 | 0.216 (0.2127) | 0.212 (0.1259) | 0.105 (0.0890) | 0.122 (0.0831)
  Eosinophils, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Eosinophils, Week 4 | 0.191 (0.2070) | 0.190 (0.0968) | 0.124 (0.0928) | 0.146 (0.0788)
  Eosinophils, Week 6: number analyzed (Participants) | 14 | 14 | 16 | 17
  Eosinophils, Week 6 | 0.202 (0.2548) | 0.229 (0.1294) | 0.134 (0.0982) | 0.150 (0.1001)
  Lymphocytes, Day 1: number analyzed (Participants) | 18 | 17 | 16 | 18
  Lymphocytes, Day 1 | 1.844 (0.5415) | 1.662 (0.4552) | 1.473 (0.6332) | 1.602 (0.7284)
  Lymphocytes, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Lymphocytes, Week 1 | 1.842 (0.7012) | 1.673 (0.5261) | 1.677 (0.7965) | 1.676 (0.4949)
  Lymphocytes, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Lymphocytes, Week 2 | 1.629 (0.4686) | 1.741 (0.5192) | 1.356 (0.5137) | 1.533 (0.4984)
  Lymphocytes, Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  Lymphocytes, Week 3 | 1.813 (0.5515) | 1.765 (0.5392) | 1.475 (0.6234) | 1.461 (0.4769)
  Lymphocytes, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Lymphocytes, Week 4 | 1.795 (0.4517) | 1.736 (0.6919) | 1.428 (0.5980) | 1.330 (0.4753)
  Lymphocytes, Week 6: number analyzed (Participants) | 14 | 14 | 16 | 17
  Lymphocytes, Week 6 | 1.739 (0.4910) | 1.491 (0.5122) | 1.427 (0.6358) | 1.466 (0.4890)
  Monocytes, Day 1: number analyzed (Participants) | 18 | 17 | 16 | 18
  Monocytes, Day 1 | 0.384 (0.1602) | 0.345 (0.1516) | 0.319 (0.1405) | 0.373 (0.1056)
  Monocytes, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Monocytes, Week 1 | 0.418 (0.1731) | 0.375 (0.1110) | 0.371 (0.1564) | 0.452 (0.1438)
  Monocytes, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Monocytes, Week 2 | 0.400 (0.2730) | 0.339 (0.1533) | 0.305 (0.1543) | 0.383 (0.1502)
  Monocytes, Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  Monocytes, Week 3 | 0.452 (0.2295) | 0.388 (0.1431) | 0.362 (0.2196) | 0.418 (0.1424)
  Monocytes, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Monocytes, Week 4 | 0.305 (0.1420) | 0.388 (0.1440) | 0.365 (0.1515) | 0.367 (0.1030)
  Monocytes, Week 6: number analyzed (Participants) | 14 | 14 | 16 | 17
  Monocytes, Week 6 | 0.369 (0.1085) | 0.336 (0.1363) | 0.350 (0.1832) | 0.430 (0.2099)
  Total Neutrophils, Day 1: number analyzed (Participants) | 18 | 17 | 16 | 18
  Total Neutrophils, Day 1 | 4.654 (2.4954) | 4.808 (1.8599) | 4.533 (1.4186) | 4.614 (1.5539)
  Total Neutrophils, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Total Neutrophils, Week 1 | 5.076 (4.0917) | 4.670 (1.4631) | 4.203 (1.1729) | 5.337 (1.8429)
  Total Neutrophils, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Total Neutrophils, Week 2 | 4.305 (2.1472) | 4.523 (1.9377) | 4.121 (1.1545) | 4.746 (1.6545)
  Total Neutrophils, Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  Total Neutrophils, Week 3 | 4.588 (1.7936) | 4.789 (1.8229) | 4.181 (1.1934) | 5.011 (2.1326)
  Total Neutrophils, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Total Neutrophils, Week 4 | 3.834 (1.4080) | 5.238 (1.8348) | 4.315 (1.5435) | 4.539 (2.1457)
  Total Neutrophils, Week 6: number analyzed (Participants) | 14 | 14 | 16 | 17
  Total Neutrophils, Week 6 | 4.163 (1.6961) | 4.061 (1.0597) | 4.126 (1.0044) | 4.891 (2.2261)
  Platelet Count, Day 1: number analyzed (Participants) | 18 | 17 | 16 | 18
  Platelet Count, Day 1 | 199.9 (67.77) | 229.9 (75.44) | 219.2 (55.11) | 223.5 (54.94)
  Platelet Count, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Platelet Count, Week 1 | 204.8 (67.74) | 219.8 (63.48) | 225.8 (57.90) | 238.8 (65.47)
  Platelet Count, Week 2: number analyzed (Participants) | 16 | 14 | 15 | 17
  Platelet Count, Week 2 | 211.3 (71.56) | 230.1 (67.64) | 209.7 (46.40) | 229.9 (70.86)
  Platelet Count, Week 3: number analyzed (Participants) | 17 | 12 | 17 | 17
  Platelet Count, Week 3 | 211.5 (71.24) | 237.3 (72.13) | 208.5 (42.24) | 224.6 (63.49)
  Platelet Count, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Platelet Count, Week 4 | 184.6 (52.35) | 255.8 (91.96) | 215.3 (52.46) | 240.5 (82.69)
  Platelet Count, Week 6: number analyzed (Participants) | 15 | 14 | 16 | 17
  Platelet Count, Week 6 | 195.1 (58.58) | 207.9 (78.54) | 217.9 (52.66) | 227.1 (68.05)
  WBC count (absolute), Day 1: number analyzed (Participants) | 18 | 17 | 16 | 18
  WBC count (absolute), Day 1 | 7.14 (2.558) | 7.06 (2.311) | 6.51 (1.570) | 6.76 (1.747)
  WBC count (absolute), Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  WBC count (absolute), Week 1 | 7.56 (4.001) | 6.92 (1.885) | 6.42 (1.740) | 7.67 (2.080)
  WBC count (absolute), Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  WBC count (absolute), Week 2 | 6.57 (2.370) | 6.84 (2.400) | 5.93 (1.099) | 6.80 (1.798)
  WBC count (absolute), Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  WBC count (absolute), Week 3 | 7.11 (1.840) | 7.18 (2.231) | 6.14 (1.275) | 7.04 (1.980)
  WBC count (absolute), Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  WBC count (absolute), Week 4 | 6.16 (1.451) | 7.57 (2.346) | 6.26 (1.617) | 6.42 (2.106)
  WBC count (absolute), Week 6: number analyzed (Participants) | 14 | 14 | 16 | 17
  WBC count (absolute), Week 6 | 6.50 (2.075) | 6.14 (1.454) | 6.06 (1.044) | 6.97 (2.327)

30. Secondary Outcome: Absolute Values of Mean Corpuscle Volume at Baseline, Week 1, 2, 3, 4 and 6
Description: Hematology parameter mean corpuscle volume was assessed at Baseline (Day 1 pre-dose), Week 2, 3, 4, and at follow-up visit (Week 6).
Time Frame: Baseline (Day 1 pre-dose), Week 1, 2, 3, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtolitre (FL)
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
Femtolitre (FL)
  Mean Corpuscle Volume, Day 1: number analyzed (Participants) | 18 | 17 | 16 | 18
  Mean Corpuscle Volume, Day 1 | 93.8 (7.29) | 92.4 (5.90) | 94.8 (5.50) | 94.2 (5.01)
  Mean Corpuscle Volume, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Mean Corpuscle Volume, Week 1 | 93.6 (7.03) | 92.7 (6.64) | 94.6 (5.97) | 95.3 (3.56)
  Mean Corpuscle Volume, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Mean Corpuscle Volume, Week 2 | 93.9 (7.34) | 92.8 (6.40) | 95.5 (5.93) | 95.4 (4.78)
  Mean Corpuscle Volume, Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  Mean Corpuscle Volume, Week 3 | 93.6 (7.47) | 93.1 (6.61) | 95.6 (5.79) | 95.9 (4.87)
  Mean Corpuscle Volume, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Mean Corpuscle Volume, Week 4 | 93.9 (7.16) | 93.4 (6.58) | 96.1 (5.92) | 95.7 (5.35)
  Mean Corpuscle Volume, Week 6: number analyzed (Participants) | 15 | 14 | 16 | 17
  Mean Corpuscle Volume, Week 6 | 94.1 (7.23) | 94.1 (4.41) | 95.8 (5.98) | 95.1 (4.81)

31. Secondary Outcome: Absolute Values of Mean Corpuscle Hgb Concentration at Baseline (Day 1), Week 1, 2, 3, 4, and 6
Description: Hematology parameter Mean Corpuscle Hgb Concentration was assessed at Baseline (Day 1 pre-dose), Week 2, 3, 4, and at follow-up visit (Week 6).
Time Frame: Baseline (Day 1 pre-dose), Week 1, 2, 3, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
G/L
  Mean Corpuscle Hgb, Day 1: number analyzed (Participants) | 18 | 17 | 16 | 18
  Mean Corpuscle Hgb, Day 1 | 328.6 (8.98) | 330.9 (5.85) | 330.2 (4.74) | 328.4 (7.87)
  Mean Corpuscle Hgb, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Mean Corpuscle Hgb, Week 1 | 329.3 (7.47) | 330.1 (7.90) | 330.8 (6.69) | 328.0 (8.46)
  Mean Corpuscle Hgb, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Mean Corpuscle Hgb, Week 2 | 327.3 (7.72) | 329.9 (6.78) | 331.3 (7.70) | 326.5 (8.61)
  Mean Corpuscle Hgb, Week 3: number analyzed (Participants) | 17 | 12 | 17 | 17
  Mean Corpuscle Hgb, Week 3 | 328.4 (5.56) | 329.5 (7.53) | 331.2 (6.12) | 326.0 (8.67)
  Mean Corpuscle Hgb, Week 4: number analyzed (Participants) | 14 | 13 | 16 | 16
  Mean Corpuscle Hgb, Week 4 | 329.6 (5.81) | 328.8 (7.83) | 329.6 (3.95) | 326.1 (7.52)
  Mean Corpuscle Hgb, Week 6: number analyzed (Participants) | 15 | 14 | 16 | 17
  Mean Corpuscle Hgb, Week 6 | 326.4 (7.36) | 330.7 (8.70) | 331.4 (5.74) | 328.2 (8.17)

32. Secondary Outcome: Absolute Values of Reticulocyte Count at Baseline (Day 1), Week 1, 2, 3, 4, and 6
Description: Hematology parameter reticulocyte were assessed at Baseline (Day 1 pre-dose), Week 2, 3, 4, and at follow-up visit (Week 6).
Time Frame: Baseline (Day 1 pre-dose), Week 1, 2, 3, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
Ratio
  Reticulocytes, Day 1: number analyzed (Participants) | 18 | 17 | 16 | 18
  Reticulocytes, Day 1 | 0.0183 (0.00584) | 0.0179 (0.00494) | 0.0208 (0.00747) | 0.0188 (0.00757)
  Reticulocytes, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Reticulocytes, Week 1 | 0.0185 (0.00667) | 0.0198 (0.00446) | 0.0256 (0.01086) | 0.0284 (0.00635)
  Reticulocytes, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Reticulocytes, Week 2 | 0.0178 (0.00558) | 0.0201 (0.00432) | 0.0224 (0.00993) | 0.0268 (0.00592)
  Reticulocytes, Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  Reticulocytes, Week 3 | 0.0191 (0.00641) | 0.0189 (0.00388) | 0.0229 (0.00943) | 0.0232 (0.00570)
  Reticulocytes, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Reticulocytes, Week 4 | 0.0174 (0.00486) | 0.0187 (0.00615) | 0.0203 (0.00905) | 0.0236 (0.00650)
  Reticulocytes, Week 6: number analyzed (Participants) | 15 | 14 | 16 | 17
  Reticulocytes, Week 6 | 0.0154 (0.00490) | 0.0196 (0.00681) | 0.0161 (0.00889) | 0.0142 (0.00700)

33. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet Count, WBC Count (Absolute) at Week 1, 2, 3, 4, and 6
Description: Baseline values were recorded on Day 1. If the Day 1 value was missing, the last non-missing value from week -1 or week-2 was represented as the baseline value. The change from baseline was calculated by subtracting the baseline value from the individual post-dose visit values. Change from Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet count, WBC count (absolute) at Week 1, 2, 3, 4, and 6 were reported.
Time Frame: Baseline (Day 1), Week 1, 2, 3, 4, and 6
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
10^9 cells/L
  Basophils, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Basophils, Week 1 | -0.000 (0.0153) | -0.011 (0.0228) | 0.008 (0.0260) | 0.003 (0.0214)
  Basophils, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Basophils, Week 2 | 0.004 (0.0145) | -0.013 (0.0300) | -0.001 (0.0202) | 0.004 (0.0336)
  Basophils, Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  Basophils, Week 3 | 0.004 (0.0229) | -0.005 (0.0273) | -0.001 (0.0218) | 0.002 (0.0221)
  Basophils, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Basophils, Week 4 | 0.005 (0.0241) | -0.000 (0.0310) | -0.003 (0.0239) | -0.001 (0.0232)
  Basophils, Week 6: number analyzed (Participants) | 14 | 14 | 16 | 17
  Basophils, Week 6 | -0.000 (0.0157) | -0.003 (0.0276) | -0.003 (0.0230) | -0.001 (0.0169)
  Eosinophils, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Eosinophils, Week 1 | -0.014 (0.0724) | -0.014 (0.0896) | -0.029 (0.0841) | 0.023 (0.0774)
  Eosinophils, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Eosinophils, Week 2 | -0.033 (0.0821) | 0.021 (0.0914) | -0.013 (0.0919) | -0.031 (0.0636)
  Eosinophils, Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  Eosinophils, Week 3 | -0.014 (0.0908) | 0.012 (0.0893) | -0.040 (0.0553) | -0.018 (0.0695)
  Eosinophils, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Eosinophils, Week 4 | -0.020 (0.0855) | -0.004 (0.0971) | -0.028 (0.0881) | 0.011 (0.0818)
  Eosinophils, Week 6: number analyzed (Participants) | 14 | 14 | 16 | 17
  Eosinophils, Week 6 | -0.012 (0.0638) | 0.034 (0.1241) | -0.018 (0.0871) | 0.009 (0.1048)
  Lymphocytes, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Lymphocytes, Week 1 | -0.002 (0.4362) | 0.024 (0.3340) | 0.126 (0.3811) | 0.048 (0.3660)
  Lymphocytes, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Lymphocytes, Week 2 | -0.234 (0.2874) | 0.062 (0.2353) | -0.176 (0.2424) | -0.036 (0.3978)
  Lymphocytes, Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  Lymphocytes, Week 3 | -0.050 (0.2860) | 0.072 (0.3048) | -0.028 (0.3650) | 0.021 (0.3838)
  Lymphocytes, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Lymphocytes, Week 4 | -0.137 (0.3011) | 0.030 (0.4575) | -0.082 (0.4047) | -0.081 (0.3471)
  Lymphocytes, Week 6: number analyzed (Participants) | 14 | 14 | 16 | 17
  Lymphocytes, Week 6 | -0.186 (0.3510) | -0.086 (0.3537) | -0.083 (0.3372) | 0.025 (0.3096)
  Monocytes, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Monocytes, Week 1 | 0.034 (0.1288) | 0.042 (0.1359) | 0.032 (0.1258) | 0.096 (0.1305)
  Monocytes, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Monocytes, Week 2 | 0.009 (0.1702) | 0.029 (0.0862) | -0.044 (0.1469) | 0.025 (0.1182)
  Monocytes, Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  Monocytes, Week 3 | 0.060 (0.1330) | 0.075 (0.0859) | 0.015 (0.1634) | 0.054 (0.1240)
  Monocytes, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Monocytes, Week 4 | -0.039 (0.1160) | 0.070 (0.0924) | 0.005 (0.1120) | -0.007 (0.1223)
  Monocytes, Week 6: number analyzed (Participants) | 14 | 14 | 16 | 17
  Monocytes, Week 6 | -0.012 (0.1245) | 0.006 (0.1212) | -0.010 (0.1160) | 0.066 (0.1579)
  Total Neutrophils, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Total Neutrophils, Week 1 | 0.422 (3.6206) | 0.027 (0.6517) | -0.362 (1.2527) | 0.457 (0.9942)
  Total Neutrophils, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Total Neutrophils, Week 2 | 0.155 (1.4350) | -0.217 (1.0644) | -0.400 (0.9470) | 0.086 (0.9817)
  Total Neutrophils, Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  Total Neutrophils, Week 3 | 0.014 (1.4591) | -0.101 (0.7464) | -0.373 (1.0319) | 0.335 (1.2442)
  Total Neutrophils, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Total Neutrophils, Week 4 | -0.394 (1.7757) | 0.493 (0.8534) | -0.239 (1.1614) | -0.148 (0.9234)
  Total Neutrophils, Week 6: number analyzed (Participants) | 14 | 14 | 16 | 17
  Total Neutrophils, Week 6 | -0.229 (1.4571) | -0.278 (0.6628) | -0.428 (1.0110) | 0.215 (1.4295)
  Platelet count, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Platelet count, Week 1 | 4.833 (21.3906) | -7.375 (23.5142) | 6.056 (31.6627) | 14.500 (19.4672)
  Platelet count, Week 2: number analyzed (Participants) | 16 | 14 | 15 | 17
  Platelet count, Week 2 | 16.375 (30.2189) | -10.500 (26.3373) | 0.200 (23.6649) | 12.941 (25.5721)
  Platelet count, Week 3: number analyzed (Participants) | 17 | 12 | 17 | 17
  Platelet count, Week 3 | 14.118 (44.4324) | -3.333 (21.8812) | -7.412 (26.8632) | 8.176 (29.1574)
  Platelet count, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Platelet count, Week 4 | -1.357 (12.9591) | 12.417 (34.3973) | -0.563 (47.3497) | 22.500 (46.0232)
  Platelet count, Week 6: number analyzed (Participants) | 15 | 14 | 16 | 17
  Platelet count, Week 6 | 8.933 (16.1973) | -14.071 (44.0742) | 2.063 (21.3868) | 10.647 (31.0764)
  WBC count (absolute), Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  WBC count (absolute), Week 1 | 0.422 (3.4155) | 0.050 (0.7598) | -0.211 (1.5885) | 0.639 (0.9960)
  WBC count (absolute), Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  WBC count (absolute), Week 2 | -0.100 (1.5786) | -0.136 (1.1972) | -0.625 (1.0866) | 0.050 (1.0377)
  WBC count (absolute), Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  WBC count (absolute), Week 3 | 0.018 (1.5653) | 0.046 (0.8373) | -0.435 (1.0571) | 0.394 (1.3908)
  WBC count (absolute), Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  WBC count (absolute), Week 4 | -0.579 (1.7494) | 0.567 (0.8659) | -0.344 (1.4846) | -0.206 (1.1174)
  WBC count (absolute), Week 6: number analyzed (Participants) | 14 | 14 | 16 | 17
  WBC count (absolute), Week 6 | -0.443 (1.5994) | -0.336 (0.8409) | -0.538 (1.0893) | 0.329 (1.4347)

34. Secondary Outcome: Change From Baseline in Mean Corpuscle Volume at Week 1, 2, 3, 4, and 6
Description: Baseline values were recorded on Day 1. If the Day 1 value was missing, the last non-missing value from week -1 or week-2 was represented as the baseline value. The change from baseline was calculated by subtracting the baseline value from the individual post-dose visit values. Change from Baseline in Mean Corpuscle Volume at Week 1, 2, 3, 4, and 6 were reported.
Time Frame: Baseline (Day 1), Week 1, 2, 3, 4, and 6
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: FL
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
FL
  Mean Corpuscle Volume, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Mean Corpuscle Volume, Week 1 | -0.222 (1.3956) | 0.125 (1.3601) | -0.222 (1.5551) | 0.278 (1.1275)
  Mean Corpuscle Volume, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Mean Corpuscle Volume, Week 2 | 0.188 (1.4705) | -0.214 (1.1217) | 0.125 (1.4549) | 0.944 (0.8726)
  Mean Corpuscle Volume, Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  Mean Corpuscle Volume, Week 3 | -0.235 (1.6405) | -0.231 (1.0127) | 0.118 (1.9327) | 1.176 (0.8828)
  Mean Corpuscle Volume, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Mean Corpuscle Volume, Week 4 | -0.143 (1.9945) | 0.083 (1.1645) | 0.188 (1.9397) | 1.188 (1.5152)
  Mean Corpuscle Volume, Week 6: number analyzed (Participants) | 15 | 14 | 16 | 17
  Mean Corpuscle Volume, Week 6 | -0.133 (1.5523) | -0.071 (1.2688) | -0.125 (2.2174) | 0.353 (1.2719)

35. Secondary Outcome: Change From Baseline in Mean Corpuscle Hgb Concentration at Week 1, 2, 3, 4, and 6
Description: Baseline values were recorded on Day 1. If the Day 1 value was missing, the last non-missing value from week -1 or week-2 was represented as the baseline value. The change from baseline was calculated by subtracting the baseline value from the individual post-dose visit values. Change from Baseline in Mean Corpuscle Hgb Concentration at Week 1, 2, 3, 4, and 6 were reported.
Time Frame: Baseline (Day 1), Week 1, 2, 3, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
G/L
  Mean Corpuscle Hgb Concentration, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 18
  Mean Corpuscle Hgb Concentration, Week 1 | 0.667 (6.9367) | -0.688 (5.3631) | 0.222 (5.8767) | -0.389 (6.3165)
  Mean Corpuscle Hgb Concentration, Week 2: number analyzed (Participants) | 16 | 14 | 16 | 18
  Mean Corpuscle Hgb Concentration, Week 2 | -0.875 (8.8835) | -0.214 (5.9249) | 0.750 (8.2341) | -2.111 (5.7792)
  Mean Corpuscle Hgb Concentration, Week 3: number analyzed (Participants) | 17 | 13 | 17 | 17
  Mean Corpuscle Hgb Concentration, Week 3 | 0.647 (7.7938) | -0.462 (6.4371) | 0.294 (8.6658) | -2.588 (8.5225)
  Mean Corpuscle Hgb Concentration, Week 4: number analyzed (Participants) | 14 | 12 | 16 | 16
  Mean Corpuscle Hgb Concentration, Week 4 | 2.429 (8.2808) | -1.417 (5.0355) | -1.375 (6.7318) | -2.625 (5.5121)
  Mean Corpuscle Hgb Concentration, Week 6: number analyzed (Participants) | 15 | 14 | 16 | 17
  Mean Corpuscle Hgb Concentration, Week 6 | -1.200 (7.1534) | -1.714 (8.3245) | 0.438 (7.8568) | -0.353 (8.1620)

36. Secondary Outcome: Absolute Values of Systolic Blood Pressure and Diastolic Blood Pressure Baseline, Week 1, Week 2, Week 3, Week 4 and Week 6
Description: Absolute values of systolic blood pressure and diastolic blood pressure Baseline (Day 1), Week 1, 2, 3, 4, and 6 as vital parameters were reported. Three measurements of systolic blood pressure and diastolic blood pressure were recorded from the participant in a supine position for at least 5 minutes (allowed enough time between measurement to completely deflate and loosen the inflatable cuff).
Time Frame: Baseline (Day 1 pre-dose), Week 1, 2, 3, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeter mercury (mmHg)
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
Millimeter mercury (mmHg)
  Systolic blood pressure, Day 1 | 132.9 (14.57) | 135.5 (13.50) | 134.0 (16.96) | 140.1 (15.50)
  Systolic blood pressure, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 19
  Systolic blood pressure, Week 1 | 132.3 (19.26) | 136.0 (17.29) | 134.6 (20.52) | 137.8 (13.29)
  Systolic blood pressure, Week 2: number analyzed (Participants) | 17 | 14 | 17 | 18
  Systolic blood pressure, Week 2 | 128.4 (12.39) | 129.4 (19.45) | 129.9 (17.18) | 139.1 (14.69)
  Systolic blood pressure, Week 3: number analyzed (Participants) | 17 | 14 | 17 | 17
  Systolic blood pressure, Week 3 | 130.2 (13.20) | 133.5 (17.28) | 133.0 (19.06) | 131.7 (12.78)
  Systolic blood pressure, Week 4: number analyzed (Participants) | 16 | 12 | 16 | 17
  Systolic blood pressure, Week 4 | 132.6 (13.94) | 133.1 (21.50) | 134.2 (14.21) | 135.4 (12.97)
  Systolic blood pressure, Week 6: number analyzed (Participants) | 16 | 16 | 16 | 17
  Systolic blood pressure, Week 6 | 134.3 (17.34) | 131.7 (19.53) | 135.0 (22.79) | 130.4 (14.10)
  Diastolic blood pressure, Day 1 | 69.9 (11.70) | 69.0 (9.48) | 68.2 (8.02) | 71.7 (10.03)
  Diastolic blood pressure, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 19
  Diastolic blood pressure, Week 1 | 66.9 (11.72) | 68.8 (10.72) | 67.4 (9.72) | 71.5 (10.04)
  Diastolic blood pressure, Week 2: number analyzed (Participants) | 17 | 14 | 17 | 18
  Diastolic blood pressure, Week 2 | 67.7 (13.04) | 68.6 (10.11) | 66.0 (8.71) | 72.7 (12.65)
  Diastolic blood pressure, Week 3: number analyzed (Participants) | 17 | 14 | 17 | 17
  Diastolic blood pressure, Week 3 | 67.7 (10.41) | 69.5 (11.39) | 66.5 (10.09) | 66.9 (11.35)
  Diastolic blood pressure, Week 4: number analyzed (Participants) | 16 | 12 | 16 | 17
  Diastolic blood pressure, Week 4 | 68.9 (12.41) | 68.2 (11.94) | 66.2 (7.24) | 68.9 (10.68)
  Diastolic blood pressure, Week 6: number analyzed (Participants) | 16 | 16 | 16 | 17
  Diastolic blood pressure, Week 6 | 70.3 (11.04) | 67.2 (8.33) | 66.6 (8.26) | 70.1 (10.43)

37. Secondary Outcome: Change From Baseline in Systolic Blood Pressure and Diastolic Blood Pressure at Week 1, 2, 3, 4, and 6
Description: Three measurements of SBP and DBP were recorded from the participant in a supine position for at least 5 minutes (allowed enough time between measurement to completely deflate and loosen the inflatable cuff). Baseline values were recorded on Day 1. If the Day 1 value was missing, the last non-missing value from week -1 or week-2 was represented as the baseline value. The change from baseline was calculated by subtracting the baseline value from the individual post-dose visit values. Change from Baseline in systolic blood pressure and diastolic blood pressure at Week 1, 2, 3, 4, and 6 were reported.
Time Frame: Baseline (Day 1 pre-dose), Week 1, 2, 3, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
mmHg
  Systolic blood pressure, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 19
  Systolic blood pressure, Week 1 | -0.519 (12.4024) | 1.167 (7.1874) | 0.565 (13.6685) | -2.368 (8.9062)
  Systolic blood pressure, Week 2: number analyzed (Participants) | 17 | 14 | 17 | 18
  Systolic blood pressure, Week 2 | -3.373 (9.6414) | -5.786 (15.4381) | -5.284 (11.6117) | 1.241 (15.2259)
  Systolic blood pressure, Week 3: number analyzed (Participants) | 17 | 14 | 17 | 17
  Systolic blood pressure, Week 3 | -1.529 (13.8349) | -1.643 (9.4312) | -2.206 (13.4641) | -5.216 (13.0309)
  Systolic blood pressure, Week 4: number analyzed (Participants) | 16 | 12 | 16 | 17
  Systolic blood pressure, Week 4 | 0.854 (10.1463) | -0.944 (13.7693) | 0.844 (9.8529) | -1.510 (14.4554)
  Systolic blood pressure, Week 6: number analyzed (Participants) | 16 | 16 | 16 | 17
  Systolic blood pressure, Week 6 | 0.125 (15.6446) | -2.458 (15.8520) | 1.656 (17.5153) | -6.451 (15.9295)
  Diastolic blood pressure, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 19
  Diastolic blood pressure, Week 1 | -3.037 (8.6409) | 0.521 (7.5933) | -0.750 (7.5737) | -0.193 (6.9711)
  Diastolic blood pressure, Week 2: number analyzed (Participants) | 17 | 14 | 17 | 18
  Diastolic blood pressure, Week 2 | -1.608 (12.0348) | -0.024 (8.0133) | -2.206 (9.0633) | 1.963 (7.1189)
  Diastolic blood pressure, Week 3: number analyzed (Participants) | 17 | 14 | 17 | 17
  Diastolic blood pressure, Week 3 | -1.647 (8.7998) | 0.857 (8.1531) | -1.755 (7.8329) | -2.627 (7.5414)
  Diastolic blood pressure, Week 4: number analyzed (Participants) | 16 | 12 | 16 | 17
  Diastolic blood pressure, Week 4 | -0.625 (5.9590) | -0.111 (8.8299) | -1.615 (7.8894) | -0.667 (7.2024)
  Diastolic blood pressure, Week 6: number analyzed (Participants) | 16 | 16 | 16 | 17
  Diastolic blood pressure, Week 6 | 1.396 (7.9807) | -1.312 (10.6795) | -1.281 (7.7741) | 0.529 (8.0830)

38. Secondary Outcome: Absolute Values of Heart Rate at Baseline (Day 1), Week 1, 2, 3, 4, and 6
Description: Absolute values of heart rate at Baseline (Day 1), Week 1, 2, 3, 4, and 6 were reported as vital parameter. Three measurements of heart rate were recorded from the participant in a supine position for at least 5 minutes (allowed enough time between measurement to completely deflate and loosen the inflatable cuff).
Time Frame: Baseline (Day 1 pre-dose), Week 1, 2, 3, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
Beats per minute
  Heart rate, Day 1 | 68.4 (10.78) | 68.4 (8.07) | 69.1 (14.58) | 67.8 (7.53)
  Heart rate, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 19
  Heart rate, Week 1 | 68.7 (10.33) | 69.5 (8.71) | 69.4 (12.89) | 69.4 (9.80)
  Heart rate, Week 2: number analyzed (Participants) | 17 | 14 | 17 | 18
  Heart rate, Week 2 | 68.9 (8.95) | 67.5 (7.60) | 66.9 (13.03) | 67.6 (11.46)
  Heart rate, Week 3: number analyzed (Participants) | 17 | 14 | 17 | 17
  Heart rate, Week 3 | 71.9 (9.92) | 69.8 (10.51) | 68.7 (14.43) | 66.9 (11.96)
  Heart rate, Week 4: number analyzed (Participants) | 16 | 12 | 16 | 17
  Heart rate, Week 4 | 67.9 (9.50) | 68.5 (9.55) | 67.9 (16.29) | 65.4 (11.97)
  Heart rate, Week 6: number analyzed (Participants) | 16 | 16 | 16 | 16
  Heart rate, Week 6 | 71.0 (10.63) | 67.6 (9.27) | 68.0 (10.55) | 68.9 (13.01)

39. Secondary Outcome: Change From Baseline in Heart Rate at Week 1, 2, 3, 4, and 6
Description: Three measurements of heart rate were recorded from the participant in a supine position for at least 5 minutes (allowed enough time between measurement to completely deflate and loosen the inflatable cuff). Baseline values were recorded on Day 1. If the Day 1 value was missing, the last non-missing value from week -1 or week-2 was represented as the baseline value. The change from baseline was calculated by subtracting the baseline value from the individual post-dose visit values. change from baseline in heart rate at Week 1, 2, 3, 4, and 6 were reported.
Time Frame: Baseline (Day 1 pre-dose), Week 1, 2, 3, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
Beats per minute
  Heart rate, Week 1: number analyzed (Participants) | 18 | 16 | 18 | 19
  Heart rate, Week 1 | 0.296 (7.1005) | 1.375 (6.9088) | 0.315 (12.5898) | 1.632 (7.1258)
  Heart rate, Week 2: number analyzed (Participants) | 17 | 14 | 17 | 18
  Heart rate, Week 2 | 0.412 (7.6771) | -1.310 (7.6051) | -1.333 (5.5777) | -0.500 (6.8716)
  Heart rate, Week 3: number analyzed (Participants) | 17 | 14 | 17 | 17
  Heart rate, Week 3 | 3.392 (8.3543) | 0.976 (8.3179) | 0.412 (6.6558) | -0.510 (6.9802)
  Heart rate, Week 4: number analyzed (Participants) | 16 | 12 | 16 | 17
  Heart rate, Week 4 | -1.167 (8.7271) | 1.111 (7.0801) | -0.500 (7.0889) | -2.020 (7.8391)
  Heart rate, Week 6: number analyzed (Participants) | 16 | 16 | 16 | 16
  Heart rate, Week 6 | 1.854 (10.9029) | -0.167 (7.7993) | -0.458 (8.2846) | 0.917 (7.5134)

40. Secondary Outcome: Absolute Electrocardiogram (ECG) Parameter Values at Baseline (Screening), Week 2, 4, and 6
Description: Full 12-lead ECGs were recorded in participants who were rested supine or seated for at least 10 minutes before each reading. All ECGs were transmitted to a central reviewer for blinded assessment. Full 12-lead ECGs were recorded on the provided ECG machine that automatically calculates heart rate, PR, QRS, QT and QTc intervals. Absolute ECG parameters including PR interval, QT interval and QRS duration values at Baseline (Screening), Week 2, 4, and 6 were reported.
Time Frame: Baseline (Screening), Week 2, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
Milliseconds (msec)
  PR Interval, Day 1: number analyzed (Participants) | 8 | 6 | 6 | 9
  PR Interval, Day 1 | 160.750 (31.1849) | 164.727 (38.0430) | 165.313 (29.3513) | 177.630 (23.4002)
  PR Interval, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 16
  PR Interval, Week 2 | 165.961 (26.2271) | 187.002 (38.5301) | 172.909 (29.4006) | 176.875 (24.4073)
  PR Interval, Week 4: number analyzed (Participants) | 15 | 13 | 16 | 15
  PR Interval, Week 4 | 161.689 (33.5960) | 180.000 (25.7034) | 174.875 (29.2025) | 176.000 (31.8927)
  PR Interval, Week 6: number analyzed (Participants) | 14 | 16 | 14 | 15
  PR Interval, Week 6 | 153.914 (19.9718) | 183.314 (42.9671) | 175.321 (32.9893) | 179.307 (31.1222)
  QRS Duration, Day 1: number analyzed (Participants) | 8 | 6 | 7 | 9
  QRS Duration, Day 1 | 99.750 (14.9833) | 101.227 (29.7471) | 99.532 (9.2023) | 106.444 (20.6101)
  QRS Duration, Week 2: number analyzed (Participants) | 17 | 15 | 18 | 18
  QRS Duration, Week 2 | 107.647 (22.2899) | 101.111 (19.1603) | 102.328 (17.8897) | 106.556 (21.4729)
  QRS Duration, Week 4: number analyzed (Participants) | 15 | 13 | 17 | 17
  QRS Duration, Week 4 | 101.467 (20.1127) | 104.205 (22.4275) | 103.965 (20.4125) | 104.392 (25.2312)
  QRS Duration, Week 6: number analyzed (Participants) | 14 | 16 | 15 | 17
  QRS Duration, Week 6 | 96.186 (14.2459) | 104.729 (21.0227) | 101.811 (18.7734) | 105.617 (22.9352)
  Uncorrected QT Interval, Day 1: number analyzed (Participants) | 8 | 6 | 7 | 9
  Uncorrected QT Interval, Day 1 | 412.000 (33.7554) | 432.455 (37.7870) | 405.541 (25.1111) | 426.074 (25.1141)
  Uncorrected QT Interval, Week 2: number analyzed (Participants) | 17 | 15 | 18 | 18
  Uncorrected QT Interval, Week 2 | 411.804 (40.7532) | 422.837 (35.0150) | 408.936 (33.1958) | 419.444 (36.1943)
  Uncorrected QT Interval, Week 4: number analyzed (Participants) | 15 | 13 | 17 | 17
  Uncorrected QT Interval, Week 4 | 413.111 (32.4499) | 413.333 (34.7435) | 411.859 (42.7345) | 423.255 (44.3408)
  Uncorrected QT Interval, Week 6: number analyzed (Participants) | 14 | 16 | 15 | 17
  Uncorrected QT Interval, Week 6 | 404.500 (34.8993) | 428.077 (34.7094) | 396.778 (32.4936) | 417.686 (45.1037)
  QTc Interval (Bazett's), Day 1: number analyzed (Participants) | 8 | 6 | 7 | 9
  QTc Interval (Bazett's), Day 1 | 430.833 (21.5149) | 446.712 (35.2019) | 435.351 (30.0154) | 437.593 (33.7848)
  QTc Interval (Bazett's), Week 2: number analyzed (Participants) | 17 | 15 | 18 | 18
  QTc Interval (Bazett's), Week 2 | 440.843 (25.7892) | 440.390 (24.2664) | 428.144 (28.4053) | 431.500 (34.3464)
  QTc Interval (Bazett's), Week 4: number analyzed (Participants) | 15 | 13 | 17 | 17
  QTc Interval (Bazett's), Week 4 | 435.556 (23.1025) | 434.590 (20.6551) | 429.480 (31.0592) | 426.549 (32.4467)
  QTc Interval (Bazett's), Week 6: number analyzed (Participants) | 14 | 16 | 15 | 17
  QTc Interval (Bazett's), Week 6 | 444.771 (23.8784) | 441.622 (24.7866) | 429.983 (30.9609) | 431.700 (34.0017)
  QTc Interval (Fridericias's), Day 1: number analyzed (Participants) | 8 | 6 | 7 | 9
  QTc Interval (Fridericias's), Day 1 | 424.417 (20.2310) | 441.424 (31.0923) | 424.970 (23.7320) | 433.815 (28.8483)
  QTc Interval (Fridericias's), Week 2: number analyzed (Participants) | 17 | 15 | 18 | 18
  QTc Interval (Fridericias's), Week 2 | 430.549 (26.2520) | 434.178 (23.6892) | 421.124 (22.9709) | 426.944 (30.0734)
  QTc Interval (Fridericias's), Week 4: number analyzed (Participants) | 15 | 13 | 17 | 17
  QTc Interval (Fridericias's), Week 4 | 427.711 (23.0747) | 427.103 (20.4117) | 422.943 (28.9082) | 424.961 (32.3172)
  QTc Interval (Fridericias's), Week 6: number analyzed (Participants) | 14 | 16 | 15 | 17
  QTc Interval (Fridericias's), Week 6 | 430.357 (22.9401) | 436.666 (22.8305) | 418.161 (24.9461) | 426.591 (33.2459)

41. Secondary Outcome: Change From Baseline in ECG Parameters at Week 2, 4 and 6
Description: Full 12-lead ECGs were recorded in participants who were rested supine or seated for at least 10 minutes before each reading. All ECGs were transmitted to a central reviewer for blinded assessment. Full 12-lead ECGs were recorded on the provided ECG machine that automatically calculates heart rate, PR, QRS, QT and QTc intervals. Baseline ECG values were defined as measurements taken at screening. The change from baseline was calculated by subtracting the baseline value from the individual post-dose visit values.
Time Frame: Baseline (Screening), Week 2, 4, and 6
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 18 | 17 | 18 | 19
msec
  PR Interval, Week 2: number analyzed (Participants) | 17 | 15 | 17 | 16
  PR Interval, Week 2 | -1.2 (9.22) | 3.6 (15.61) | 2.5 (9.88) | -0.6 (10.80)
  PR Interval, Week 4: number analyzed (Participants) | 15 | 13 | 16 | 15
  PR Interval, Week 4 | -2.6 (17.37) | 1.8 (9.97) | 3.1 (12.35) | -2.0 (16.16)
  PR Interval, Week 6: number analyzed (Participants) | 14 | 16 | 14 | 15
  PR Interval, Week 6 | -5.8 (10.70) | 0.5 (16.22) | -0.2 (16.83) | 1.3 (15.67)
  QRS Duration, Week 2: number analyzed (Participants) | 17 | 15 | 18 | 18
  QRS Duration, Week 2 | 2.5 (7.69) | -0.0 (5.80) | 0.4 (7.29) | 4.6 (4.94)
  QRS Duration, Week 4: number analyzed (Participants) | 15 | 13 | 17 | 17
  QRS Duration, Week 4 | -0.4 (13.82) | 1.8 (4.80) | 1.3 (5.32) | 2.3 (8.15)
  QRS Duration, Week 6: number analyzed (Participants) | 14 | 16 | 15 | 17
  QRS Duration, Week 6 | -0.3 (8.07) | 0.2 (10.04) | -1.9 (6.64) | 3.5 (5.07)
  Uncorrected QT Interval, Week 2: number analyzed (Participants) | 17 | 15 | 18 | 18
  Uncorrected QT Interval, Week 2 | -10.8 (28.14) | -1.9 (12.25) | 3.1 (15.31) | 5.8 (22.23)
  Uncorrected QT Interval, Week 4: number analyzed (Participants) | 15 | 13 | 17 | 17
  Uncorrected QT Interval, Week 4 | -2.9 (21.31) | -10.9 (18.75) | 5.4 (17.87) | 8.8 (20.89)
  Uncorrected QT Interval, Week 6: number analyzed (Participants) | 14 | 16 | 15 | 17
  Uncorrected QT Interval, Week 6 | -7.9 (20.94) | -2.4 (17.34) | -6.7 (15.39) | 3.2 (31.45)
  QTc Interval (Bazett's), Week 2: number analyzed (Participants) | 17 | 15 | 18 | 18
  QTc Interval (Bazett's), Week 2 | 7.9 (18.96) | 3.4 (11.28) | -4.0 (12.98) | 1.7 (17.77)
  QTc Interval (Bazett's), Week 4: number analyzed (Participants) | 15 | 13 | 17 | 17
  QTc Interval (Bazett's), Week 4 | 2.5 (15.30) | -0.8 (10.26) | -1.8 (14.87) | -1.9 (19.04)
  QTc Interval (Bazett's), Week 6: number analyzed (Participants) | 14 | 16 | 15 | 17
  QTc Interval (Bazett's), Week 6 | 11.4 (17.49) | 2.9 (12.94) | 0.0 (20.99) | 3.3 (19.38)
  QTc Interval (Fridericias's), Week 2: number analyzed (Participants) | 17 | 15 | 18 | 18
  QTc Interval (Fridericias's), Week 2 | 1.6 (12.03) | 1.7 (7.80) | -1.7 (10.68) | 3.0 (17.12)
  QTc Interval (Fridericias's), Week 4: number analyzed (Participants) | 15 | 13 | 17 | 17
  QTc Interval (Fridericias's), Week 4 | 1.0 (11.26) | -4.2 (10.16) | 0.5 (13.54) | 1.6 (17.45)
  QTc Interval (Fridericias's), Week 6: number analyzed (Participants) | 14 | 16 | 15 | 17
  QTc Interval (Fridericias's), Week 6 | 4.6 (12.04) | 1.0 (11.36) | -2.4 (15.05) | 3.2 (18.08)

42. Secondary Outcome: Mean Maximum Plasma Concentration (Cmax) of GSK1278863 and GSK1278863 Metabolites
Description: Cmax of GSK1278863 and GSK1278863 metabolites (M1, M2, M3, M4, M5 and M6) were reported. For assessment of Pharmacokinetics parameters blood samples were collected at Day 1 (pre-dose), Week 2 (first samples was collected approximately between 4 to 8 h and then 1, 2 and 3 h after this first sample) and Week 4 (Pre-dose 1, 2 and 3 h post-dose).
Time Frame: Day 1 (pre-dose), Week 2 (first samples was collected approximately between 4 to 8 h and then 1, 2 and 3 h after this first sample) and Week 4 (Pre-dose 1, 2 and 3 h post-dose).
Population: All participants from whom a pharmacokinetic sample had been obtained and analyzed were included in the pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Arm/Group | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 13 | 17 | 18
nanogram per millilitre (ng/mL)
  GSK1278863 | 2.68 (92.6) | 12.8 (121) | 35.7 (143)
  M2 | 1.03 (27.9) | 3.83 (61.4) | 10.3 (61.1)
  M3 | 1.23 (25.1) | 4.45 (54.4) | 11.8 (64.8)
  M4 | 0.721 (29.7) | 2.74 (84.7) | 7.29 (116)
  M5 | 0.296 (23.7) | 1.08 (49.0) | 2.81 (79.8)
  M6 | 0.455 (21.9) | 1.74 (56.1) | 4.43 (83.1)

43. Secondary Outcome: Mean Steady State Area Under the Curve (AUC) of GSK1278863 and GSK1278863 Metabolites
Description: Mean Steady state AUC of GSK1278863 and GSK1278863 metabolites (M1, M2, M3, M4, M5 and M6) were reported. For pharmacokinetic parameter assessment blood samples were collected at Day 1 (pre-dose), Week 2 (first samples was collected approximately between 4 to 8 h and then 1, 2 and 3 h after this fist sample) and Week 4 (Pre-dose 1, 2 and 3 h post-dose).
Time Frame: as for outcome 42
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
Number analyzed (Participants) | 13 | 17 | 18
ng*hour/mL
  GSK1278863 | 10.3 (119) | 51.1 (159) | 148 (167)
  M2 | 13.0 (38.8) | 51.9 (81.3) | 140 (65.4)
  M3 | 17.8 (33.4) | 67.1 (74.2) | 175 (71.6)
  M4 | 5.54 (60.0) | 22.0 (99.0) | 63.4 (105)
  M5 | 4.64 (27.7) | 17.3 (66.7) | 43.5 (86.0)
  M6 | 5.34 (36.3) | 21.5 (71.4) | 56.3 (85.8)

ADVERSE EVENTS:
Time Frame: Up to follow up contact (Week 6).
Description: Safety population was used for analysis of SAEs and nSAEs.
Arm/Group | Placebo | GSK1278863, 0.5 mg | GSK1278863, 2 mg | GSK1278863, 5 mg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17 | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/17 | 2/18 | 1/19
Other Adverse Events (participants affected / at risk) | 8/18 | 10/17 | 5/18 | 5/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | GSK1278863, 0.5 mg (N=17) | GSK1278863, 2 mg (N=18) | GSK1278863, 5 mg (N=19)
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | GSK1278863, 0.5 mg (N=17) | GSK1278863, 2 mg (N=18) | GSK1278863, 5 mg (N=19)
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Conduction disorder (Cardiac disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.